



## **Statistical Analysis Plan (SAP)**

**Protocol title:** An Open-Label Extension Study to Evaluate Long-

Term Efficacy and Safety of A4250 in Children with Progressive Familial Intrahepatic Cholestasis Types 1

and 2 (PEDFIC 2)

**Protocol no.:** A4250-008

**IND no:** 130591

**EudraCT no.:** 2017-002325-38

**Protocol version no., date:** Amendment 06, 21 Dec 2021

**Document version no., date:** Final v2.1, 04 Apr 2024

**Prepared by:** Firma Clinical Research





## Signature Page

| Prep | ared by: | DDD | |
|------|---------------------------|-------------------|------|
| F | PPD | PPD<br>Signature: | |
| | Firma Clinical Research | Email: | |
| | Tillia Cillicai Rescarcii | | Data |
| | | Signature | Date |
| Revi | ewed by: | DDD | |
| | PPD | PPD<br>Signature: | |
| | Firma Clinical Research | Email: | |
| | | Signature | Date |
| Revi | ewed and approved by: | PPD | |
| | PPD | Signature: | |
| | IPSEN Pharmaceuticals | Email: | |
| | II SEIVI haimaccaicais | | |
| | DDD | Signature | Date |
| | PPD | PPD | |
| | | Signature: | |
| | IPSEN Pharmaceuticals. | Email: | |
| | | Signature | Date |





## **Revision History**

| VERSION/DATE | MODIFIED BY | REASON FOR MODIFICATIONS |
|---|---|---|
| Final v1.0/20Mar2020 | NA | |
| Final v1.1/11Aug2020 | PPD | To clarify missing data will not be imputed for analysis. |
| | | 2. To update dictionary version. |
| | | 3. To clarify the growth analysis will be based on derived growth data using the software or methods from the Centers for Disease Control and Prevention (CDC) website for patients with age ≥ 2 years old and from the WHO website for patients with age < 2 years old. |
| | | <ul><li>4. To clarify the counting of number of adverse events.</li><li>5. To clarify that local laboratory data will be used when central laboratory data are not available.</li></ul> |
| | | 6. To clarify the calculation of change from baseline for AM&PM pruritus scores (daily, weekly, bi-weekly, monthly) for analysis purposes. |
| | | 7. To update the analysis windows of non-<br>eDiary assessments. |
| | | 8. To add the analysis windows for the endpoints of eDiary assessments. |
| Final v1.2/25Aug2020 | PPD | To clarify the baseline derivation of serum bile acid |
| Final v2.0/22Aug2022 | PPD | To add BRIC patients per protocol amendment 06 |
| | | 2. Dose regimen can be initiated with 40 or 120 µg/kg/day |
| | | 3. Add additional interim analysis (IA) |





| VERSION/DATE | MODIFIED BY | REASON FOR MODIFICATIONS |
|---|---|---|
| Final v2.1/04Apr2024 | PPD | To add header sample for final CSR tables. |
| | | <ol><li>To update endpoints to add the visit<br/>during extension period if available.</li></ol> |
| | | <ol><li>To update the analysis windows for<br/>patient entering extension period.</li></ol> |
| | | 4. To follow the criteria for liver monitoring per protocol amendment 06. |
| | | 5. To update disposition categories. |
| | | <ol><li>To update the definition of TEAE by<br/>adding "Within 28 days follow-up after the<br/>last dose of odevixibat".</li></ol> |
| | | <ol> <li>To update the rule for laboratory related<br/>efficacy endpoints to only consider the data<br/>up to 14 days follow up after the last dose of<br/>odevixibat.</li> </ol> |
| | | 8. To add analysis of change from baseline 1 and 2 for serum bile acid, pruritus, and growth. Baseline 1 is only for odevixibat treated patients in Cohort 1. |
| | | <ol><li>To add proportion of responders for<br/>pruritus scores as secondary endpoint.</li></ol> |
| | | 10. To add change and shift in use of UDCA and/or Rifampicin at Weeks 24, 48, and 72 in secondary endpoint. |
| | | 11. To add listing for BRIC patients for<br>episodic flares during the study treatment in<br>exploratory endpoint. |
| | | 12. To add any possible sequelae of FSV deficiency TEAEs by SOC and PT. |
| | | 13. To add PT Terms of possible sequelae of FSV deficiency into Appendix G. |





# **Table of Contents**

| Signature Page | 2 |
|---|---|
| Revision History | 3 |
| Table of Contents | 5 |
| List of Appendices | 7 |
| List of Tables. | 7 |
| List of Figures | 8 |
| List of Abbreviations | 9 |
| 1. Introduction | 12 |
| 2. Study Objectives | 12 |
| 2.1 Primary Objectives | 12 |
| 2.2 Secondary Objectives | 13 |
| 3. Study Design | 13 |
| 3.1 General Study Design | 13 |
| 3.2 Randomisation and Blinding | 18 |
| 3.3 Study Treatments and Assessments | 18 |
| 3.3.1 Serum Bile Acids | 19 |
| 3.3.2 Itching, Scratching, and Sleep Score | 20 |
| 3.3.3 Growth | 20 |
| 3.3.4 Biomarker Sample | 21 |
| 3.3.5 Change of Antipruritic Medication | 21 |
| 3.3.6 Quality of Life Questionnaire (PedsQL) | 21 |
| 3.3.7 PELD/MELD Score | 21 |
| 3.3.8 Fibroscan <sup>®</sup> | 22 |
| 3.3.9 Markers of Fibrosis | 23 |
| 3.3.10 Liver Biopsy | 23 |
| 3.3.11 Global Impression of Change and Global Impression of Symptom Measures | |
| 4. Study Endpoints | |
| 4.1 Primary Efficacy Endpoints | |





| | 4.2 | Secondary Efficacy Endpoints | 25 |
|---|---|---|---|
| | 4.3 | Exploratory Endpoints | 27 |
| | 4.4 | Safety Evaluation | 29 |
| 5. | S | ample Size and Power | 30 |
| 6. | Iı | nterim Analysis | 30 |
| 7. | A | Analysis Sets | 31 |
| 8. | S | tatistical Considerations and Analysis | 31 |
| | 8.1 | Handling of Missing Data and/or Invalid Data and Outliers | 31 |
| | 8. | 1.1 Missing Data Analysis Methods for Efficacy Endpoints | 31 |
| 9. | S | tatistical Methods | 31 |
| | 9.1 | General Statistical Conventions | 31 |
| | 9.2 | Patient Disposition | 33 |
| | 9.3 | Protocol Deviations | 34 |
| | 9.4 | Demographic and Baseline Characteristics | 34 |
| | 9.4.1 | 1 Demographic Characteristics | 34 |
| | 9.4 | 4.2 Baseline and Disease Characteristics | 35 |
| | 9.4 | 4.3 Medical and Surgical History | 36 |
| | 9.4 | 4.4 Prior and Concomitant Medications | 36 |
| | 9.5 | Extent of Exposure | 37 |
| | 9.: | 5.1 Treatment Duration. | 37 |
| | 9.: | 5.2 Treatment Compliance | 38 |
| | | 9.5.2.1 Source Data from CRFs | 38 |
| | | 9.5.2.2 Source Data from eDiary | 38 |
| | 9.6 | Efficacy Analyses | 39 |
| | 9. | 6.1 Analysis Methods | 39 |
| | 9. | 6.2 Treatment by Centre Interaction Analysis (Multicentre Study) | 39 |
| | 9. | 6.3 Analyses of Primary Efficacy Endpoints | 39 |
| | 9. | 6.4 Analyses of Secondary Endpoints | 40 |
| | 9.0 | 6.5 Analyses of Exploratory Endpoints | 43 |
| | 9.7 | Safety Analyses | 45 |





| 9.7.1 | Adverse Events | 45 |
|---|---|---|
| | Definition for TEAEs of Fat-Soluble Vitamin Deficiency, bea, and Hepatotoxicity | 48 |
| 9.7.1.2 | Definitions and Determination of Hepatic Events | 49 |
| 9.7.2 | Clinical Laboratory Evaluations | 52 |
| 9.7.3 | Vital Sign Measurements | 54 |
| 9.7.4 | Physical Examinations | 54 |
| 9.8 Other | r Analyses | 55 |
| 9.8.1 | Subgroup Analyses | 55 |
| 9.8.2 | Data Safety Monitoring Board | 55 |
| 10. Changes | to Planned Analysis from Study Protocol | 55 |
| 11. Appendi | ces | 57 |
| List of Appen | dices | |
| Appendix A: | Derived Variables | 57 |
| Appendix B: | Visit Window | 62 |
| Appendix C: | Definition of Region Variable | 67 |
| Appendix D: | Handling of Missing or Incomplete Dates | 68 |
| Appendix E: | Normal Reference Ranges of Vital Signs | 70 |
| Appendix F: | SI and US Conventional Units of Clinical Laboratory Values | 72 |
| Appendix G: | PT Term of Possible Sequelae of FSV Deficiency | 73 |
| List of Tables | | |
| Table 1: Fibro | scan Scoring for Cholestatic Liver Disease (Fibrosis Score) | 23 |
| Table 2: Contr | rolled Attenuation Parameter Score and Steatosis Grading | 23 |
| Table 3: Deriv | ved Variables for Demographic and Baseline Characteristics, Various Duration Derivations, Drug Compliance, Baseline Derivations, and Other Important Derivations | |
| Table 4: Analy | ysis Visit Window (General) | 62 |
| Table 5: Analy | ysis Visit Windows for GIC/GIS, Physical Measurements and Selected Lab Test) | 63 |





Version v2.1; Date: 04Apr2024 

| Table 6: Ana | lysis Visit Window for PedsQL, Fibroscan, Abdominal Ultrasound and AFP | 64 |
|---|---|---|
| Table 7: Ana | lysis Visit Window for eDiary Parameters | 65 |
| Table 8: Ana | lysis Visit Window for Proportion of Responders for Pruritus Monthly Scores | 66 |
| Table 9: Ana | lysis Visit Window for Proportion of Responders for Pruritus Bi-<br>weekly Scores | 66 |
| Table 10: An | alysis Visit Window for Proportion of Positive Pruritus Assessment | 67 |
| Table 11: De | finition of Region Variable | 68 |
| Table 12: He | art Rate by Age (Beats/Minute) Reference | 70 |
| Table 13: No | ormal Respiratory Rate by Age (Breaths/Minute) Reference | 70 |
| Table 14: No | ormal Blood Pressure by Age (mm Hg) Reference | 70 |
| Table 15: No | rmal Temperature Range by Method | 71 |
| List of Figur | es | |
| Figure 1 | Study Design | 16 |
| Figure 2 | Study Design for Cohort 2 as of Protocol Amendment 6 | 16 |





## List of Abbreviations

| <b>Abbreviation</b> | <u>Definition</u> |
|---------------------|----------------------------------------------------|
| AE(s) | Adverse Event(s) |
| AFP | Alfa-fetoprotein |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| APRI | Aspartate Aminotransferase to Platelet Ratio Index |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BRIC | Benign Recurrent Intrahepatic Cholestasis |
| CAP | Controlled Attenuation Parameter |
| CDC | Centers for Disease Control and Prevention |
| CDF | Cumulative Distribution Function |
| CI | Confidence Interval |
| COVID-19 | Coronavirus Disease 2019 |
| CPK | Creatine Phosphokinase |
| CSR | Clinical Study Report |
| DSMB | Data Safety and Monitoring Board |
| eCRF | Electronic Case Report Form |
| eDiary | Electronic Diary |
| EOT | End of Treatment |
| EU | European Union |
| FAS | Full Analysis Set |
| Fib-4 | Fibrosis-4 |
| GGT | Gamma-glutamyl Transferase |
| GIC | Global Impression of Change |
| GIS | Global Impression of Symptoms |

Informed Consent Form

ICF





**Abbreviation Definition** 

ICH International Council for Harmonisation

INR international normalised ratio

ISE Integrated Summary of Effectiveness

ISS Integrated Summary of Safety

LDH Lactate Dehydrogenase

MAA Marketing Authorisation Application

MedDRA Medical Dictionary for Regulatory Activities

MELD Model for End-stage Liver Disease

NA Not Applicable

NAPPED Natural Course and Prognosis of PFIC and Effect of biliary

Diversion

NDA New Drug Application

ObsRO Observer-reported Outcome

p-C4 Plasma 7α-hydroxy-4-cholesten-3-one Concentration

PedsQL Pediatric Quality of Life Inventory
PELD Paediatric End-stage Liver Disease

PFIC Progressive Familial Intrahepatic Cholestasis

PRO Patient-reported Outcome

PT Preferred Term

QoL Quality of Life

RoW Rest of World

SAE(s) Serious Adverse Event(s) SAP Statistical Analysis Plan

SAS® Statistical Analysis System Software

SE Standard Error

SI International System of Unit

SOC System Organ Class
StdDev Standard Deviation
T Telephone Contact





| <b>Abbreviation</b> | <b>Definition</b> |
|---------------------|-------------------------------------|
| TEAE(s) | Treatment-emergent Adverse Event(s) |
| TFLs | Tables, Figures, and Listings |
| ULN | Upper Limit of Normal |
| US | United States |
| V | Clinic Visit |
| VS | Visit Screening |
| WHO | World Health Organization |





#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to provide detailed descriptions of the statistical methods, data derivations, and data displays for Study Protocol A4250-008, An Open-Label Extension Study to Evaluate Long-Term Efficacy and Safety of A4250 in Children with Progressive Familial Intrahepatic Cholestasis Types 1 and 2 (PEDFIC 2). The table of contents and templates for the tables, figures, and listings (TFLs) will be produced in a separate document.

Any deviations from this SAP will be described and justified in the clinical study report (CSR). The preparation of this SAP has been based on International Council for Harmonisation (ICH) E3 and E9 guidelines<sup>1</sup>,<sup>2</sup>. All data analyses and generation of TFLs will be performed using Statistical Analysis System (SAS®) software (Version 9.4 or higher). The SAP will be finalised and signed off prior to locking the database.

#### 2. Study Objectives

## 2.1 Primary Objectives

#### Cohort 1

To demonstrate a sustained effect of odevixibat (A4250) on serum bile acids and pruritus in children with progressive familial intrahepatic cholestasis (PFIC) Types 1 and 2.

#### Cohort 2

To evaluate the effect of odevixibat on serum bile acids and pruritus in patients with PFIC who either (1) Do not meet eligibility criteria for Study A4250-005 (PEDFIC 1) or (2) Patients who do meet the eligibility criteria for Study A4250-005 after recruitment of Study A4250-005 has been completed.

<sup>&</sup>lt;sup>1</sup> ICH Topic E3: Structure and Content of Clinical Study Reports (CPMP/ICH/137/95- adopted December 1995)

<sup>&</sup>lt;sup>2</sup> ICH Topic E9: Statistical Principles for Clinical Trials (CPMP/ICH/363/96 – adopted March 1998).





## 2.2 Secondary Objectives

#### Cohorts 1 and 2:

- To evaluate the long-term safety and tolerability of repeated daily doses of odevixibat
- To evaluate the effect of odevixibat on growth
- To evaluate the effect of odevixibat on biliary diversion and/or liver transplantation
- To evaluate the effect of odevixibat on biochemical markers of cholestasis and liver disease

## 3. Study Design

#### 3.1 General Study Design

This is a Phase 3, multicentre, open-label extension study to investigate the long-term efficacy and safety of odevixibat at doses of 40 and 120 µg/kg/day in patients with PFIC, including episodic forms also referred to as benign recurrent intrahepatic cholestasis (BRIC). Cohort 1 includes children with PFIC Types 1 and 2 who have participated in Study A4250-005. Cohort 2 includes patients with any type of PFIC who have elevated serum bile acids and cholestatic pruritus and who either (1) did not meet eligibility criteria for Study A4250-005 (PEDFIC 1) or (2) were eligible for enrolment in Study A4250-005 after recruitment of Study A4250-005 completed. Up to 40 patients' post-biliary diversion surgery were allowed to participate in Cohort 2.

Study data are reviewed periodically (approximately on a quarterly basis) by a Data Safety and Monitoring Board (DSMB) until the last patient reaches 72 weeks.

Informed consent must have been obtained before any study procedures were performed. After signing the informed consent form (ICF), patients were evaluated for study eligibility and considered to be enrolled in the study. For Cohort 1, patients were eligible to participate in this extension study if they completed the 24 weeks of treatment in Study A4250-005, or, prior to amendment 6 of the A4250-005 protocol, withdrew from Study A4250-005 after a minimum of 12 weeks of treatment with odevixibat due to





patient/caregiver judgment of no improvement/intolerable symptoms but met all inclusion criteria and no exclusion criteria. Patients who withdrew from Study A4250-005 due to a study drug-related adverse event (AE) were not eligible. For Cohort 2, patients meeting all inclusion criteria and no exclusion criteria were eligible.

Before protocol amendment 6 of the A4250-008 protocol, eligible patients were enrolled into this open-label extension study and treated with a daily dose of odevixibat 120 μg/kg/day for 72 weeks. Patients not tolerating the 120 μg/kg/day dose after a minimum of 1 week had the option to down-titrate to a lower dose (40 µg/kg/day). The patient was to return to the higher dose as soon as deemed appropriate by the investigator. Under protocol amendment 6, patients entering Cohort 2 were to start treatment at 40 μg/kg/day with the possibility to dose escalate to 120 μg/kg/day after 12 weeks if there was no improvement in pruritus based on investigator judgment. The patient could return to the lower dose if the 120 µg/kg/day dose was not tolerated following a minimum of 1 week of treatment. Any dose titration was to be done in consultation with the sponsor Medical Monitor or designee. Patients who wished to continue receiving odevixibat after 72 weeks had the option to remain on treatment in an extension period with visits every 16 weeks until the drug was commercially available, provided continued use was supported by the risk-benefit profile and the patient had not been previously withdrawn or discontinued from the study. In that case the 4-week Follow-up period would not occur.

Patients in Cohort 2 went through a Screening period consisting of 2 clinic visits as follows:

- Visit S-1: Screening Visit 1 (Days -56 to -35)
- Visit S-2: Screening Visit 2 (Days -28 to -7)

Patients who did not meet eligibility criteria may have been re-screened after consultation with the Medical Monitor. Patients not fulfilling inclusion/exclusion criteria after 3 attempts were not allowed to rescreen.

All patients were to have a minimum of 12 clinic visits and 6 scheduled telephone contacts (see Figure 1 and Figure 2) as follows:





- Visit 1: Screening/inclusion visit (Day 1; coincided with Visit 9/End of Treatment (EOT) in Study A4250-005 for patients in Cohort 1. Assessments that were performed at Visit 9/EOT during Study A4250-005 were not to be repeated.)
- Visit 2: Week 4
  - Telephone contact 1: Week 8
- Visit 3: Week 12
  - Telephone contact 2: Week 18
- Visit 4: Week 22
- Visit 5: Week 24
  - Telephone contact 3: Week 30
- Visit 6: Week 36
  - Telephone contact 4: Week 42
- Visit 7: Week 46
- Visit 8: Week 48
  - Telephone contact 5: Week 54
- Visit 9: Week 60
  - Telephone contact 6: Week 66
- Visit 10: Week 70
- Visit 11: Week 72/optional extension period
- Visit 12: Follow-up visit; Week 76 (for those not participating in optional extension period)
- Optional extension period visits every 16 weeks; Week 88 and onwards





Figure 1 Study Design



QD: once daily; T: telephone contact; V: study visit; VS: Visit Screening

Note: Visit 1 coincides with Visit 9 of Study A4250-005. Patients who are not tolerating the 120 µg/kg/day dose may be down-titrated to the 40 µg/kg/day dose following a minimum of 1 week of treatment. The patient can return to the higher dose as soon as deemed appropriate.

This figure is only applicable to Cohort 2 up to Protocol Amendment 5. Figure 2 presents the study design for Cohort 2 as of Protocol Amendment 6.

Figure 2 Study Design for Cohort 2 as of Protocol Amendment 6



QD: once daily; T: telephone contact; V: study visit; VS: Visit Screening

Note: As of Protocol Amendment 6, patients entering Cohort 2 will start treatment at 40 µg/kg/day with the possibility to dose escalate to 120 µg/kg/day after 12 weeks if there is no improvement in pruritus based on investigator judgment. The patient can return to the lower dose if the 120 µg/kg/day dose is not tolerated following a minimum of 1 week of treatment.

Patients were to return to the clinic at Weeks 4 and 12 and thereafter every 10 to 12 weeks for follow-up measurements. Between clinic visits there was to be a telephone contact with the patient and/or caregiver to report AEs. Additional clinic visits may have been required for patients who needed direct site assistance for AE monitoring for safety maintenance and other assessments.

At Visit 11, patients were to be offered the choice to continue receiving odevixibat treatment in an optional extension period. During the optional extension period the patient was to receive odevixibat at the same dose as at the end of the 72-week treatment





period, returning to the clinic every 16 weeks until the drug is commercially available, provided continued use was supported by the risk-benefit profile and the patient had not been previously withdrawn or discontinued from study.

If a patient was prematurely withdrawn from the study prior to Week 72, all assessments scheduled for Visit 11 were to be performed at the time the patient withdrew. If a patient participating in the optional extension study withdrew prior to commercial drug availability, all assessments scheduled for the optional extension period EOT visit were to be performed.

If a liver biopsy was performed according to the local regulations or standard of care at any time during A4250-008, the biopsy results should have been recorded in the electronic case report form (eCRF). If liver biopsy results were collected for a patient in Study A4250-005 or prior to Week 24 in Study A4250-008, the patient was to be asked to consent to a follow-up liver biopsy at Visit 11, if allowed per local regulations, unless 2 prior liver biopsy results had been collected (with at least 1 year between biopsies). Liver biopsies were not performed in Spain.

For patients not participating in the optional extension period, Visit 12 was to take place 28 days after Visit 11. All patients who were prematurely withdrawn were to have this visit 28 days after the last dose of study drug for AE monitoring and other safety follow-up assessments.

If a patient discontinued before Week 72, additional telephone contacts were to be made every 3 months after the Follow-up visit (Visit 12) up to Week 72 to inquire whether the patient had undergone biliary diversion or liver transplantation, and if ongoing TEAEs at the time of discontinuation had resolved. The telephone calls were to take place up until 72 weeks even if the patient had biliary diversion or liver transplant.

Patients and/or caregivers were instructed to complete the electronic diary (eDiary) every morning and evening for the first 24 weeks (Visits 1 to 5) and for the 21 days before each clinic visit thereafter (Visits 6 to 12). In addition, Cohort 2 patients and/or caregivers were instructed to complete the eDiary during the Screening period. Patients participating in the optional extension period were not to complete eDiary entries after Visit 11. The eDiary included patient-reported outcome (PRO) and observer reported outcome (ObsRO) items for evaluation of itching (using PRO), scratching (using ObsRO), and





sleep disturbance (using both PRO and ObsRO). ObsRO in patients of all ages was recorded by a caregiver. If possible, the same caregiver was to complete the ObsRO items throughout the study. Additionally, caregivers were requested to report in the diary the time that study drug was administered during the treatment period.

The study nurse was to monitor eDiary compliance by routine review of the CRF Health website. If both diary entries were missing on a specific day during this time, the study nurse was to call the caregiver/patient with a reminder to complete all scheduled entries. Non-compliance was to be documented and explained in the source documents.

## 3.2 Randomisation and Blinding

Not applicable (NA).

#### 3.3 Study Treatments and Assessments

Prior to Amendment 6 of the protocol, all patients were dosed with 120  $\mu$ g/kg/day for 72 weeks. As of Amendment 6, patients enrolled in Cohort 2 received 40  $\mu$ g/kg/day for at least the first 12 weeks with the option to increase the dose to 120  $\mu$ g/kg/day for the remaining 60 weeks if there was no improvement in pruritus based on investigator judgement. Patients not tolerating the 120  $\mu$ g/kg/day dose after a minimum of 1 week for reasons other than new liver findings and severe diarrhoea had the option to down-titrate to a lower dose (40  $\mu$ g/kg/day). They were to return to the higher dose as soon as deemed appropriate by the Investigator. More than one upward dose titration (from 40  $\mu$ g/kg/day directly to 120  $\mu$ g/kg/day) for the same event was not recommended. If, in the opinion of the Investigator, a dose titration should be considered prior to the 1-week minimum, the Investigator was to consult with the Medical Monitor or designee. Any dose titration should have been done in consultation with the Sponsor Medical Monitor or designee.

Study drug was to be dispensed to the patient at defined intervals from Visit 1 through Visit 9, together with instructions on how to store and take the drug. Study drug administration data, including whether each patient took each dose or partial doses of study drug, whether there were any delayed or missed doses, and whether the capsule was opened or swallowed whole, was to be documented through the diaries and transferred to the study database.





Patients participating in the optional extension period were to continue at the same dose as at the end of the 72-week treatment period ( $120 \,\mu g/kg/day$  or  $40 \,\mu g/kg/day$ ). Patients not tolerating the dose at any time throughout the extension period were to have the option to down-titrate to a lower dose ( $40 \,\mu g/kg/day$ ) following consultation with the Sponsor Medical Monitor or designee. Patients were to return to the higher dose as soon as deemed appropriate by the Investigator. More than one upward dose titration (from  $40 \,\mu g/kg/day$ ) directly to  $120 \,\mu g/kg/day$ ) for the same event was not recommended.

Bottles with 34 capsules were to be given to the patient at each visit. A patient who required 2 or more capsules per day was to be given multiple bottles; please refer to the investigational product manual. If a patient's weight changed at any time during the study, dose adjustment was required. The number of capsules provided to the patient was to be based on the body weight thresholds identified in Protocol A4250-008, Table 3.

Odevixibat was to be taken in the morning together with food. On clinic visits days when laboratory assessments were conducted (Visits 1 to 10; and every 16 weeks thereafter for those participating in the optional extension period), study drug was to be taken after the visit.

Efficacy assessments and daily recording of pruritus using an eDiary in this study are briefly introduced as follows.

#### 3.3.1 Serum Bile Acids

Blood samples for analysis of fasting total serum bile acids were to be drawn at all visits from Visit 1 (Visit S-1 for Cohort 2) through Visit 12. Fasting serum bile acids were also to be drawn at all visits (every 16 weeks) during the optional extension period. Patients were to fast (water intake only) for at least 4 hours prior to the collection of samples for serum bile acids. Exceptions could be made for infants <12 months of age if unable to fast for the full 4 hours. For any visit at which a bile acid sample result was unreportable, an additional unscheduled visit for a repeat sample collection may have been scheduled. Samples were to be handled and transported to a central laboratory per instructions in the laboratory manual.





#### 3.3.2 Itching, Scratching, and Sleep Score

Itching, observed scratching, and sleep disturbance were to be recorded twice each day via the eDiary. Patient and/or caregivers were instructed to fill in the eDiary every morning (AM score representing nighttime itching/scratching and sleep disturbance) and evening (PM score representing daytime itching/scratching and tiredness) for the first 24 weeks and the last 21 days before all the remaining visits to the clinic. There was to be no interruption between Visits 11 and 12. Patients participating in the optional extension period stopped eDiary entries at Visit 11. Patients and/or caregivers were instructed to complete the eDiary in the morning after the patient awakened and in the evening just before the patient went to sleep.

The eDiary includes Albireo ObsRO and PRO items. Patients <8 years of age were not asked to complete the Albireo PRO items; the Albireo ObsRO was to be completed by caregivers of patients in this age group. Older patients, ≥ 8 years of age, completed the Albireo PRO items and the caregiver completed the Albireo ObsRO items. The Albireo PRO items assess severity of itch, aspects of sleep disturbance (morning diary only), and tiredness. For patients 8 to 12 years of age, the caregiver read the Albireo PRO items along with the child and recorded the child's response. A guide was provided to the caregivers that provided standardised explanations of the Albireo PRO items, in case the patient was confused or required clarification about the meaning of a question. The Albireo ObsRO items assess severity of observed scratching, aspects of observed sleep disturbance (morning diary only), and observed signs of tiredness (evening diary only). The Albireo ObsRO and PRO scratching and itch severity items use 0 to 4 response scales, where each response is distinguished by a unique facial expression, verbal anchor, number, and colour code.

#### **3.3.3** Growth

Prior to Amendment 6 of the protocol, standard height measurements were obtained, and weight was evaluated using a certified weight scale. As of Amendment 6, growth (height and weight) was to be measured by the standardized assessments outlined in the US FDA guidance document, Orally Inhaled and Intranasal Corticosteroids: Evaluation of the Effects on Growth in Children (March 2007). Height and length (velocity) was to be





measured using a certified stadiometer and weight (Z-score) using a certified weight scale.

Mid-arm circumference (3 repeat measurements) was to be collected at the study site for all patients after Protocol Amendment 6.

Study sites were trained on using a standardized approach when measuring height with a stadiometer and additional detailed instructions were provided in study documents.

BMI was calculated by weight (kg) / height (m)<sup>2</sup>. Change was defined as linear growth deficit (weight and BMI for age) compared to a standard growth curve.

## 3.3.4 Biomarker Sample

Blood samples for plasma  $7\alpha$ -hydroxy-4-cholesten-3-one concentration (p-C4) and autotaxin were to be drawn at Visits 1, 2, 5, 8, and 11 for patients with body weight >10 kg. Samples were to be handled and transported to a central laboratory per instructions in the laboratory manual.

## 3.3.5 Change of Antipruritic Medication

Any change of antipruritic medication must be noted in the eCRF.

## 3.3.6 Quality of Life Questionnaire (PedsQL)

Patients and caregivers were asked to complete a quality of life (QoL) questionnaire, the Pediatric Quality of Life Inventory (PedsQL), at Visits 1, 5, 8, 11 and at all visits of the optional extension period. Details of the questions included on the questionnaire are located in Appendix 4 of the protocol.

#### 3.3.7 PELD/MELD Score

The paediatric end-stage liver disease (PELD) score was calculated for children under 12 years of age. For children 12 years of age or older, the model for end-stage liver disease (MELD) score was calculated.





For calculation of the PELD/MELD score<sup>3</sup> laboratory parameters will be converted in following units:

- Total bilirubin in mg/dL
- Albumin in g/dL
- Creatinine in mg/dL

PELD score =  $4.80 * \ln(\text{total bilirubin}) + 18.57 * \ln(\text{INR}) - 6.87 * \ln(\text{albumin}) + 4.36 (if patient <1 year: scores for patients listed for liver transplantation before the patient's first birthday continue to include the value assigned for age (<1 year) until the patient reaches the age of 24 months) + 6.67 (if the patient has growth failure [< -2 StdDev])$ 

Laboratory values <1.0 were set to 1.0 for the calculation of the PELD score.

MELD score = 9.57 \* ln(creatinine) + 3.78 \* ln(total bilirubin) + 11.2 \* ln(INR) + 6.43

Laboratory values <1.0 were set to 1.0 and serum creatinine values >4.0 mg/dL (equivalent of 353.6  $\mu$ mol/L) were set to 4.0 for calculation of the MELD score.

If a patient went from 11 years of age to 12 between the beginning and end of study, both PELD and MELD scores were to be calculated at the first visit after the 12th birthday and move to MELD score.

#### 3.3.8 Fibroscan®

Where available, Fibroscan® was to be performed as per institution standard practice at Visits 1, 5, 8, and 11. The data collected on the Fibroscan form (liver stiffness measured in kPa and controlled attenuation parameter (CAP) measured in dB/m) was to be

-

<sup>&</sup>lt;sup>3</sup> https://www.unos.org/wp-content/uploads/unos/MELD\_PELD\_Calculator\_Documentation.pdf; accessed on 25-Jul-2018.





converted to determine stage of fibrosis and grade of steatosis, respectively, using a score card<sup>4,5</sup> as outlined in Table 1 and Table 2.

Table 1: Fibroscan Scoring for Cholestatic Liver Disease (Fibrosis Score)

| SCORE | F0 TO F1<br>NO SCARRING/<br>MILD FIBROSIS | F2<br>MODERATE<br>FIBROSIS | F3<br>SEVERE<br>FIBROSIS | F4<br>CIRRHOSIS OR<br>ADVANCED<br>FIBROSIS |
|---|---|---|---|---|
| Fibroscan result | 2 to 7 kPa | >7 to 9 kPa | >9 to 17 kPa | >17 kPa |

Table 2: Controlled Attenuation Parameter Score and Steatosis Grading

| CONTROLLED ATTENUATION PARAMETER SCORE | AMOUNT OF LIVER WITH FATTY CHANGE | STEATOSIS GRADE |
|---|---|---|
| <238 dB/m | _ | S0 |
| 238 to 260 dB/m | 11% to 33% | S1 |
| 260 to 290 dB/m | 34% to 66% | S2 |
| >290 dB/m | ≥67% | S3 |

#### 3.3.9 Markers of Fibrosis

Aspartate aminotransferase to platelet ratio index (APRI) score and fibrosis-4 (Fib-4) score were calculated at Visits 1, 3, 5, 8, and 11.

APRI = [(AST in U/L)/(AST upper limited of normal (ULN) in U/L)]  $\times$  100/(platelets in 10<sup>9</sup>/L)

Fib-4 score = (age\*AST in U/L)/(platelets in  $10^9/L * \sqrt{(ALT in U/L)}$ ).

### 3.3.10 Liver Biopsy

If a liver biopsy was performed according to the local regulations or standard of care at any time during Study A4250-008, the biopsy results should have been recorded in the

Statistical Analysis Plan Protocol A4250-008 Version v2.1; Date: 04Apr2024 

<sup>&</sup>lt;sup>4</sup> Understanding your Fibroscan Results. Memorial Sloan-Kettering Cancer Center Web site. https://www.mskcc.org/cancer-care/patient-education/understanding-your-fibroscan-results Updated February 27, 2018. Accessed March 27, 2020.

<sup>&</sup>lt;sup>5</sup> Jewish Hospital Fibroscan Interpretation Assessment SOP. Washington University, Louisville Kentucky. https://louisville.edu/medicine/departments/medicine/divisions/gimedicine/physician-resources/calculators-and-tools-files/fibroscan-interpretation-sheet. Undated.





eCRF. If the patient had liver biopsy results collected in Study A4250-005 or prior to Week 24 in Study A4250-008, the patient was to be asked to consent to a follow-up liver biopsy, if allowed per local regulations, at Visit 11 unless 2 prior liver biopsy results had been collected with at least one year between biopsies. Liver biopsies were not performed in Spain.

# 3.3.11 Global Impression of Change and Global Impression of Symptom Measures

Patients, caregivers, and clinicians were to complete the global impression of change (GIC) and the global impression of symptom (GIS) measures at Visits 1, 2, 3, 5, 8, and 11, and at all visits during the optional extension period.

The GIC items assess change in itch (patient version), scratching (caregiver and clinician versions), and sleep (all versions) since starting the study drug. The GIS items assess itch (patient version), scratching (caregiver and clinician versions), and sleep (all versions) in the past week. Caregivers and clinicians were to complete the GIC and GIS for all patients; only patients  $\geq 8$  years of age were to complete the patient version.

A detailed description of procedures and assessments to be conducted during this study is summarised in the Table 1 Schedule of Assessments (Screening Period through Follow-up Period) and Table 2 schedule of study assessments (Optional Extension Period) of the protocol.

### 4. Study Endpoints

## 4.1 Primary Efficacy Endpoints

The primary efficacy endpoints are as follows:

• EU and Rest of the World (RoW): Change from baseline in fasting serum bile acids after 72 weeks of treatment.

Change from baseline will be calculated based on the average of the values at Weeks 70 and 72. The baseline fasting serum bile acids value is defined as follows unless otherwise specified:





Cohort 1: The average of the last 2 values before the first dose of study drug in Study A4250-008. In general, these 2 values are the values of the last 2 assessments of Study A4250-005. If pre-dose assessments are collected in Study A4250-008 for a patient, then the values of pre-dose assessments in Study A4250-008 will be considered first and used to calculate the baseline. These 2 values need to be taken from 2 consecutive scheduled visits or unscheduled visits. If only one value is available from 2 consecutive scheduled visits or unscheduled visits, then that value will be used as baseline.

Cohort 2: The average of the last 2 values before the first dose of study drug in Study A4250-008.

• United States (US): Proportion of positive pruritus assessments at the patient level over the 72-week treatment period using the Albireo ObsRO instrument.

A positive pruritus assessment is defined as a scratching score of  $\leq 1$  or at least a one-point decrease from baseline on the Albireo ObsRO instrument. At each assessment, the AM score will be compared to the baseline AM average, and the PM score will be compared to the baseline PM average. Both AM and PM pruritus assessments will be included in the analysis of this endpoint. AM scores from the period of 14 days before or on the first dose day in Study A4250-008 will be averaged as the AM baseline. PM scores from the period of 14 days before the first dose day in Study A4250-008 will be averaged as the PM baseline. If a patient's baseline average score is  $\leq 1$ , then only the criterion of a one-point drop from baseline on the Albireo ObsRO instrument will be used to determine whether a pruritus assessment is positive or not for the primary endpoint analysis.

#### 4.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints include the following:

- **EU and RoW:** Proportion of positive pruritus assessments at the patient level over the 72-week treatment period using the Albireo ObsRO instrument.
- US: Change from baseline in fasting serum bile acids after 72 weeks of treatment.
- All Regions:





- Change from baseline in serum bile acids at Weeks 4, 12, 22, 24, 36, 46, 48, 60, 70, 72, 76 and all visits (every 16 weeks) during the optional extension period.
- o Proportion of individual assessments meeting the definition of a positive pruritus assessment at the patient level using the Albireo ObsRO instrument from Weeks 0-4, Weeks 0-12, Weeks 0-22, Weeks 0-24, Weeks 0-36, Weeks 0-46, Weeks 0-48, Weeks 0-60, and Weeks 0-70, and the proportion of positive pruritus assessments at each 4--week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76.
- O Proportion of individual AM assessments meeting the definition of a positive pruritus assessment at the patient level using the Albireo ObsRO instrument from Weeks 0-4, Weeks 0-12, Weeks 0-22, Weeks 0-24, Weeks 0-36, Weeks 0-46, Weeks 0-48, Weeks 0-60, Weeks 0-70, and Weeks 0-72, and the proportion of positive pruritus assessments at each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76.
- O Proportion of individual PM assessments meeting the definition of a positive pruritus assessment at the patient level using the Albireo ObsRO instrument from Weeks 0-4, Weeks 0-12, Weeks 0-22, Weeks 0-24, Weeks 0-36, Weeks 0-46, Weeks 0-48, Weeks 0-60, Weeks 0-70, and Weeks 0-72, and the proportion of positive pruritus assessments at each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76.
- Number of patients undergoing biliary diversion surgery or liver transplantation. These parameters will be evaluated separately and together at Weeks 24, 48, 72 and all visits (every 16 weeks) during the optional extension period.
- Change in growth from baseline to Weeks 12, 24, 36, 48, 60, 72 and all
  visits (every 16 weeks) during the optional extension period after initiation
  of odevixibat treatment, defined as the linear growth deficit (height/length





for age, weight for age, and BMI) compared to a standard growth curve (Z-score, StdDev from the fiftieth percentile, P50).

- Change in APRI score and Fib-4 score from baseline to Week 72 and all visits (every 16 weeks) during the optional extension period.
- Change in PELD/MELD score from baseline to Week 72 and all visits (every 16 weeks) during the optional extension period.
- o Change in use of UDCA and/or Rifampicin at Weeks 24, 48, and 72.
- Proportion of responders for pruritus scores using the Albireo ObsRO instruments by visit (proportion of patients achieving meaningful reduction based on the clinically meaningful threshold of 1.0 point, which is estimated from the distribution-based and anchor-based approaches in the blinded psychometric analysis)

### 4.3 Exploratory Endpoints

All Exploratory Endpoints will be evaluated at Weeks 24, 48, and 72 unless otherwise noted. For summary purposes, if not otherwise specified, the baseline value of a parameter is defined as the last non-missing assessment of that parameter before the first dose of odevixibat in Study A4250-008. Exploratory efficacy endpoints include the following:

- Change in serum alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), and total bilirubin concentration from baseline to Week 72 and all visits (every 16 weeks) during the optional extension period.
- Proportion of individual assessments meeting the definition of a positive pruritus assessment at the patient level over the 72-week treatment period. A positive pruritus assessment includes an itch score ≤1, or at least a 1 -point decrease from baseline based on the Albireo PRO instrument; only patients ≥8 years of age will complete the Albireo PRO instrument.
- Change from baseline in sleep parameters by each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between





Visit 5/Week 24 and Visit 11/Week 72 over the 72-week treatment period measured with the Albireo PRO and ObsRO instruments.

- Change from baseline in international normalised ratio (INR), albumin, liver enzymes, leukocytes, and platelets from baseline to Week 72 and all visits (every 16 weeks) during the optional extension period.
- Change from baseline to all visits where assessed in measures of bile acid synthesis (autotaxin, p-C4)
- Assessment of global symptom relief at Weeks 4, 12, 24, 48, 72 and all visits (every 16 weeks) during the optional extension period as measured by patient, caregiver, and clinician GIC items.
- Change from baseline by each 4-week interval between Visit 1/Screening and
  Visit 5/Week 24, then by each visit between Visit 5/Week 24 and
  Visit 12/Week 76 in patient-reported and observer-reported night-time itching and
  scratching severity scores.
- Change from baseline by week interval from Baseline to Week 72 in patient-reported and observer-reported night-time itching and scratching severity scores.
- Change from baseline by each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76 in patient-reported and observer-reported morning time itching and scratching severity scores.
- Change from baseline by week interval from Baseline to Week 72 in observerreported morning time itching and scratching severity scores.
- Change from baseline by each 4-week interval between Visit 1/Screening and
  Visit 5/Week 24, then by each visit between Visit 5/Week 24 and
  Visit 12/Week 76 in pooled pruritus score including observer-reported scratching
  for patients <8 years of age and patient-reported itch severity for patients ≥8 years
  of age.</li>





- Change from baseline by week interval from Baseline to Week 72 in pooled pruritus score including observer-reported scratching for patients <8 years of age and patient-reported itch severity for patients ≥8 years of age.
- Change from baseline in additional patient-reported and observer-reported sleep parameters (e.g. tiredness, number of awakenings) by each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76.
- Change from baseline in PedsQL questionnaire from Baseline to Week 72 and all visits (every 16 weeks) during the optional extension period.
- Change from baseline in stage of liver fibrosis as assessed by Fibroscan® (where available).
- Change from baseline in stage of liver fibrosis, as assessed by post-treatment biopsy (when available).

## 4.4 Safety Evaluation

Safety criteria are as follows:

- The primary safety analysis for this study will include the incidence of total treatment-emergent adverse events (TEAEs) and TEAEs categorised by causality, severity, and seriousness assessments made by the Investigator.
- Trends in safety will also be evaluated for the following:
  - Physical examinations
  - Concomitant medications
  - Vital signs
  - Laboratory test results (including clinical chemistry, haematology, urinalysis, alfa-fetoprotein [AFP], vitamins A and E, 25-hydroxy vitamin D, and INR)
  - Abdominal ultrasound
  - Discontinuations due to AEs





#### 5. Sample Size and Power

There is no formal hypothesis testing in this open-label study. The sample size for Cohort 1 was determined in Study A4250-005. For Cohort 1, patients will be enrolled after completion of Study A4250-005 or participation of 12 weeks in that study. For the other endpoints, mainly descriptive analyses will be performed.

The proportion of patients with at least 1 event (i.e., surgical bile diversion, liver transplantation, death) that can be expected in a non-treated population depends on PFIC type and age distribution of the included patients. The expected proportion of patients with events will be calculated for the study population once each patient's age and PFIC type are known, using the probability that a patient will get an event estimated from the reference population in the ongoing observational cohort study, NAtural Course and Prognosis of PFIC and Effect of Biliary Diversion (NAPPED).

As an example, if the expected proportion of patients with at least 1 event is estimated to be 30% in the study population, and then if the proportion of patients with at least 1 event during odevixibat long-term treatment is shown to be only 10% in the study, the power is approximately 89% to 96% (1-sided test, alpha=2.5%) for a confidence interval (CI) with upper boundary <30% based on a sample size of n=48 to 60. The sample size of 60 for Cohort 2 was estimated based on the availability of target patient population to evaluate the therapeutic benefit for those patients.

## 6. Interim Analysis

This study is an extension study of Study A4250-005 and was ongoing at the time of the New Drug Application (NDA) and Marketing Authorisation Application (MAA) submission in November 2020. For the NDA/MAA submission purposes, the database was locked on 31Aug2020 for Study A4250-005, and an interim analysis of Study A4250-008 with data cut on 15Jul 2020 was performed to accompany the final analyses of Study A4250-005.

For this interim analysis submitted in the NDA/MAA, the analyses described in this SAP were conducted, as appropriate, based on data available at the time of the data cut-off date. The interim analysis was conducted for both safety and efficacy mainly based on descriptive statistics. The main time point was at the end of 24-week treatment period





while all data were included for by-visit summaries. These analyses accompanied the Study A4250-005 analyses and provided further information regarding the safety and efficacy of odevixibat dosing for more than 24 weeks.

For supporting a post-marketing commitment, an interim analysis of Study A4250-008 (planned data cut of 31July2022) was performed in order to update the CSR. The selected analyses described in this SAP were conducted, as appropriate, for the interim analysis based on data available at the time of the data cut-off date. The interim analysis was conducted for both safety and efficacy mainly based on descriptive statistics.

Analyses may be performed at select time points throughout the collection of patient data for regulatory requirements and sponsor decision making purposes.

## 7. Analysis Sets

The FAS will consist of all patients who received at least 1 dose of study drug in Study A4250-008. The FAS will be the primary analysis set for all analyses unless otherwise specified.

#### 8. Statistical Considerations and Analysis

### 8.1 Handling of Missing Data and/or Invalid Data and Outliers

#### 8.1.1 Missing Data Analysis Methods for Efficacy Endpoints

No imputation will be made for any missing data. The assessments after intercurrent events (death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) or follow-up assessments ( $\geq$  last dose day + 15 days) will be excluded from analysis with the exception of the analysis of patients undergoing biliary diversion surgery or liver transplantation. For eDiary data analysis, data after last dose will be excluded from analysis.

#### 9. Statistical Methods

#### 9.1 General Statistical Conventions

Study data will be reviewed periodically (approximately on a quarterly basis) by a DSMB. For DSMB analyses, the Adjudication Process Document outlines the events that





will be adjudicated and see Section 9.8.2. Descriptive statistics are mainly used in this open-label extension study unless otherwise specified. All statistical procedures will be completed using SAS®, Version 9.4 or higher.

Continuous variables will be summarised using descriptive statistics, including the number of patients with non-missing value (n), mean, median, StdDev (or standard error [SE]), minimum, and maximum. The letter "n" will be presented without a decimal point. Minimum and maximum values will be presented to the same precision as in the database. Mean and median will be presented to 1 more decimal place than the minimum and maximum. StdDev or SE will be presented to 1 more decimal place than the mean and median.

For categorical variables, summaries will include counts of patients (frequencies) and percentages. Percentages will be rounded to 1 decimal place. Descriptive summaries of change from baseline in categorical variables will be provided using shift tables, as applicable.

For summary purposes, if not otherwise specified, the baseline value of a parameter is defined as the last non-missing assessment of that parameter before the first dose of odevixibat in Study A4250-008 (Appendix A). Derived variables used for the analyses are provided in Appendix A.

Analysis windows defined in Appendix B will be applied for all laboratory parameters, questionnaires, vital sign measurements, physical examinations, and other efficacy parameters in the study, unless otherwise specified.

For the final CSR, all summaries will be presented for the following treatment groups, unless otherwise specified.

- Placebo (A4250-005) to Odevixibat (A4250-008)
- Odevixibat 40 or 120 μg/kg/day (A4250-005) to Odevixibat 120 μg/kg/day (A4250-008)
- Cohort 2 (A4250-008)
- Odevixibat Overall

Table header will be presented as follows:





| Placebo/Odevixibat <sup>a</sup> | Odevixibat/Odevixibat <sup>b</sup> | Cohort 2 <sup>c</sup> | Odevixibat |
|---|---|---|---|
| (A4250-005/A4250-008) | (A4250-005/A4250-008) | (A4250-008) | Overall |

- a Includes patients who received placebo in Study A4250-005 and transitioned to odevixibat 120 μg/kg/day in Study A4250-008
- b Includes patients who received odevixibat 40 or 120 µg/kg/day in Study A4250-005 and transitioned to odevixibat 120 µg/kg/day in Study A4250-008
- c Includes patients who received odevixibat in Cohort 2 of Study A4250-008

All patient data, including derived data, will be presented in individual patient data listings. All listings will be sorted by cohort/treatment subgroup, patient number, date/time, and visit. The sex and age for each patient will be stated on each listing. Data listings will be based on all enrolled patients.

Patients who didn't directly rollover from Study A4250-005 but enrolled in Study A4250-008 after a gap in dosing or re-enrolled in Study A4250-008 after a gap in dosing were assigned separate patient IDs. They will be considered as separate patients in all analyses.

## 9.2 Patient Disposition

All patients who provided informed consent will be included in a summary of patient accountability.

The following categories will be summarised by cohort/treatment subgroup and overall as follows:

- Patients screened
- Screening failures
- Patients eligible to receive dose
- Patients dosed
- Patients completing 72 weeks treatment period
  - o Patients not enrolled in optional extension treatment period
  - o Patients enrolled in the optional extension treatment period
    - Patients ongoing in optional extension treatment period





- Patients discontinuing optional extension treatment period (including reasons for treatment discontinuation)
- Patients discontinuing 72 weeks treatment period early (including reasons for treatment discontinuation)
- Patients who have undergone biliary diversion surgery
- Patients who have undergone liver transplantation
- Patients who have been listed for liver transplantation

Additionally, analysis populations will be summarised overall and by region (Appendix C).

#### 9.3 Protocol Deviations

All protocol deviations will be reviewed at the final protocol deviations review meeting before final database lock, through clinical input provided by the Sponsor, using the following sources of information:

• Protocol deviation logs, provided by ICON Clinical, Pharmacovigilance, Medical, and Data Management.

Important protocol deviations that are likely to impact the efficacy and safety will be identified by the study team during the manual review at the data review meeting prior to DB lock. The list of important protocol deviations will be finalized after the data review meeting. The number of patients with important protocol deviations (overall and by deviation) will be summarised by cohort/treatment subgroup and overall.

#### 9.4 Demographic and Baseline Characteristics

## 9.4.1 Demographic Characteristics

Age, height, weight, and BMI at baseline and other demographic variables, e.g. age category (<6 months, 6 months to 5 years, 6 to 12 years, 13 to 18 years, and >18 years), sex, race, ethnicity, country, region (Appendix C) will be summarised descriptively by cohort/treatment subgroup and overall.

Demographics data for Cohort 1 will be obtained from Study A4250-005, as appropriate.





#### 9.4.2 Baseline and Disease Characteristics

The following disease characteristics will be summarised by cohort/treatment subgroup and overall: years since PFIC diagnosis; type of PFIC; Bile Salt Export Pump (BSEP) subtype for PFIC 2 Patients and BSEP genotype; presence of significant pruritus per Investigator report; at least 1 serum bile acid level >100 µmol/L within 6 months before Screening visit; serum bile acid category; reasons for discontinuation of historical PFIC-related investigational medications; baseline Z-score; Use of UDCA or/and Rifampicin and diagnostic genetic laboratory test as well as Child-Pugh classification and hepatic impairment classification per NCI Organ Dysfunction Working Group.

Child-Pugh classification: mild (Class A), moderate (Class B), or severe hepatic impairment (Class C) is based on the FDA Guidance for Pharmacokinetics in Patients with Impaired Hepatic Function. Determination of the classification is made based on medical review of baseline laboratory data and medical history.

Hepatic impairment will also be classified per the NCI Organ Dysfunction Working Group classification as mild, moderate or severe (Mansfield et al. 2016)<sup>6</sup>. Both the Child-Pugh and NCI classification will be included in the baseline characteristics and both will be applied in the subgroup analysis based on hepatic impairment status.

The following continuous parameters will also be summarized: estimated glomerular filtration rate (eGFR); baseline Z-score (weight, height, BMI and mid-arm circumference); and baseline values of alanine aminotransferase (ALT); aspartate aminotransferase (AST); gamma-glutamyl transferase (GGT); total bilirubin; alkaline phosphatase; INR; and vitamins A, E, and 25 hydroxy D.

eGFR will be calculated based on the modified/bedside Schwartz equation. For patients <18 year of age, Bedside Schwartz Equation will be used:

GFR (mL/min/1.73 m<sup>2</sup>) =  $(36.2 \times \text{Height in cm}) / \text{Creatinine in } \mu \text{mol/L}$ 

For patients ≥ 18 years, the isotope dilution mass spectrometry (IDMS)-traceable Modification of Diet in Renal Disease (MDRD) Study equation will be used:

Statistical Analysis Plan Protocol A4250-008

Version v2.1; Date: 04Apr2024 

<sup>&</sup>lt;sup>6</sup> Aaron S. Mansfield, Michelle A. Rudek, Diana Vulih, Gary L. Smith, Pamela Jo Harris, and S. Percy Ivy (2016). "The effect of hepatic impairment on outcomes in phase 1 clinical trials in cancer subjects".





GFR (mL/min/1.73 m<sup>2</sup>) = 175 × (Creatinine in  $\mu$ mol/L/88.4)<sup>-1.154</sup> × (Age)<sup>-0.203</sup> × (0.742 if female) × (1.212 if African American)

The average of three repeat measurements of mid-arm circumference will be calculated for the analyses.

If length instead of height is measured for patients, height of the patients will be calculated from length by using the formula:

Height (cm) = Length (cm) -0.7 cm.

A listing will present demographic and baseline characteristics by patient. In addition, an individual listing of liver biopsy results, including historical liver biopsy results for patients in Cohort 2, will be produced.

The results of pathologic variants identified for ATP8B1, ABCB11, ABCB4, or other genes (such as NR1H4, TJP2, DCDC2, CLDN1, MYO5B) will be listed for all patients.

## 9.4.3 Medical and Surgical History

The frequencies and percentages of patients with reported medical and surgical history will be presented by system organ class (SOC) and preferred term (PT). Medical and surgical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA), Version 26.0 or later. The summary table will be sorted alphabetically by SOC and PT. Medical and surgical history will also be listed.

For patients with BRIC, a flare/cholestatic episode can be self-reported or clinically assessed based on medical history. The frequency, duration, and severity of flares within the last 6 months at a minimum, and within the last 5 years, other clinical signs and symptoms during a cholestatic episode/flare including nausea, vomiting and pruritus followed by jaundice, fatigue, weight loss, malaise, steatorrhoea, night blindness, increased bilirubin and alkaline phosphatase levels and increased INR, ALT, AST and GGT, if possible, will be listed.

## 9.4.4 Prior and Concomitant Medications

Prior and concomitant medications used in this study will be coded using the March 2023 version or later of the World Health Organisation (WHO) Drug Global Dictionary.




**Prior medication:** A medication taken by a patient within 3 months before the first dose date of study drug with a recorded medication stop date before the first dose date of study drug is a prior medication. This will not include historical PFIC-related investigational medications collected separately on CRFs.

**Concomitant medication:** A medication taken by a patient the day on or after the first dose date of study drug or a medication with a start date before the first dose date of study drug without a recorded stop date before the first dose date of study drug is a concomitant medication.

As patients in Cohort 1 enter the study directly from Study A4250-005, the summary of prior medications is provided only for Cohort 2. Concomitant medication use during the study will be summarised descriptively using frequency tables by Anatomical Therapeutic Chemical (ATC) Class 4 and PT by cohort/treatment subgroup and overall for the FAS. ATC class and PT will be presented alphabetically. All prior and concomitant medications will be listed. Details for imputing missing or partial start and/or stop dates of non-study medications are located in Appendix D.

#### 9.5 Extent of Exposure

#### 9.5.1 Treatment Duration

Exposure will be summarised with descriptive statistics (n, mean, StdDev, minimum, median, and maximum) and presented by cohort/treatment subgroup and overall.

For Cohort 2 patients who dose escalate from 40 µg/kg/day to 120 µg/kg/day, exposure at each dose and overall will be calculated.

Categorical summaries of treatment duration will also be provided. Study drug exposure will be derived as follows:

Duration of exposure (in weeks) = (date of last study drug intake – date of first study drug intake + 1)/7.

Investigators are allowed to interrupt the study drug to allow for the resolution of AEs, if necessary. Drug interruptions will not be considered when calculating treatment duration.





#### 9.5.2 Treatment Compliance

Treatment compliance will be assessed by maintaining adequate study drug dispensing records. Treatment compliance over the treatment period will be calculated using 2 sources of data.

#### 9.5.2.1 Source Data from CRFs

Treatment compliance =  $100 \times [(number of capsules dispensed - number of capsules returned)/number of capsules that should have been taken].$ 

The number of capsules that should have been taken is calculated as the number of days that patient was in the treatment period (exposure as above) multiplied by the number of prescribed capsules to be taken (based on patient's body weight, Protocol Table 3) during the treatment period. The total number of capsules actually taken is the total number of capsules recorded as taken based on the CRF (number of capsules dispensed minus returned) summed over the treatment period. If the number of capsules returned is confirmed as missing and the study drug is confirmed has not been returned, the derivation will not be done.

# 9.5.2.2 Source Data from eDiary

Treatment compliance  $=100 \times (\text{total number of capsules taken/total number of capsules planned to be taken)}$ . The number of capsules planned to be taken will be estimated based on patient's body weight per Protocol Table 3. The compliance rate based on eDiary data will be calculated during the first 24 weeks only.

The calculated compliance rates will be summarised and the one based on CRFs will be considered the primary compliance rate. The compliance rates reported by visit on the CRFs also will be summarised.

Descriptive summary statistics will be used to summarise study drug compliance by cohort and overall. The number and percentage of patients with a compliance <80%, between 80% and 120%, and >120% will also be presented.





#### 9.6 Efficacy Analyses

This section addresses the analyses to be conducted on the primary, secondary, and exploratory efficacy variables.

The efficacy analysis will be carried out using the patients from the FAS. Figures for selected efficacy endpoints, such as the primary pruritus endpoint, change in serum bile acids, and change in other patient-reported and caregiver-reported outcomes, will be provided by cohort/treatment subgroup and by visit. Forest plots will be provided for the efficacy subgroup analyses.

For efficacy endpoints derived from central laboratory data, if central laboratory data are not available due to COVID-19 or other reasons, local laboratory data will be used and converted to standard unit used by central laboratory. In addition, laboratory related efficacy endpoints will only be considered up to 14 days follow-up after the last dose.

#### 9.6.1 Analysis Methods

Descriptive statistics mainly will be used in this open-label extension study unless otherwise specified.

#### 9.6.2 Treatment by Centre Interaction Analysis (Multicentre Study)

NA

#### 9.6.3 Analyses of Primary Efficacy Endpoints

All the primary analyses will be based on the FAS, unless otherwise specified.

For the EU and RoW, change from baseline 2 in fasting serum bile acids will be analysed by using the 1-sample t-test or the Wilcoxon signed rank test, as appropriate at the end of the 72-week treatment period based on the average of the values at Weeks 70 and 72. Baseline 2, defined in the table of derived variables in Appendix A, will be used to calculate change from baseline for the summary.

For Cohort 1 patients who were on odevixibat in Study A4250-005, change from Baseline 1 to end of the 72-week treatment in Study A4250-008 will be analysed by using the 1-sample t-test or the Wilcoxon signed rank test, as appropriate. Baseline 1,





defined in the table of derived variables in Appendix A, will be used for this statistical analysis.

For the US, the proportion of positive pruritus assessments at the patient level over the 72-week treatment period using the Albireo ObsRO instrument will be summarised descriptively. A positive pruritus assessment is defined as a scratching score of ≤1 or at least a 1-point drop from baseline on the Albireo ObsRO instrument. At each assessment, the AM score will be compared to the baseline AM average, and the PM score will be compared to the baseline PM average. Both AM and PM pruritus assessments will be included in the analysis of this endpoint. For analysis purposes, diary entries will be assigned to a study day based on the recorded date regardless of recorded time. AM scores from the period of 14 days before or on the first dose day in Study A4250-008 will be averaged as AM baseline. PM scores from the period of 14 days before the first dose day in Study A4250-008 will be averaged as PM baseline. If a patient's baseline score is ≤1, then only the criterion of a one-point drop from baseline on the Albireo ObsRO instrument will be used to determine whether a pruritus assessment is positive or not for the primary endpoint analysis. Rounded baseline score will be used for the analysis.

A 95% CI will be provided for the proportion of positive pruritus assessments.

Change from Baseline 1 and 2 in monthly scratching severity score to end of the 72-week treatment in Study A4250-008 will be analysed by using the 1-sample t-test or the Wilcoxon signed rank test, as appropriate. Baseline 1 will only be used for patients in Cohort 1 who were on odevixibat in Study A4250-005.

# 9.6.4 Analyses of Secondary Endpoints

All secondary analyses will primarily be summarised descriptively based on the FAS, unless otherwise specified.

The change in secondary endpoints such as serum bile acids, growth, APRI score, Fib-4 score, PELD/MELD will be summarised by visit using descriptive statistics.

#### Growth

Change in growth (height/length for age, weight for age, mid-arm circumference for age, and BMI for age) will be analysed by using the 1-sample t-test or the Wilcoxon signed





rank test, as appropriate at the end of the 72-week treatment period based on the average of the values at Weeks 70 and 72. In addition, change in growth will also be displayed using graphical presentations. Baseline 1 and 2, defined in the table of derived variables in Appendix A, will be used to calculate change from baseline for data analysis. Baseline 1 will only be used for patients in Cohort 1 who were on odevixibat in Study A4250-005.

The analysis of growth data for height/length, weight, and BMI will be based on calculated values using the software or methods from the Centers for Disease Control and Prevention (CDC) website for patients with age  $\geq 2$  years old and from the WHO website for patients with age  $\leq 2$  years old<sup>7,8</sup>. The analysis of growth data for mid-arm circumference will be based on calculated values for 2 months to 18 years for U.S. Children<sup>9</sup>. CRF collected growth data will be listed.

#### Serum Bile Acids

For serum bile acids assessments, if a patient has assessments at Weeks 70 and 72, then the average of the 2 assessment values at Weeks 70 and 72 will be used for data analysis. This handling will also be applied to Weeks 22 and 24, and Weeks 46 and 48.

# Proportion of Positive Pruritus

The proportion of individual assessments meeting the definition of a positive pruritus assessment at the patient level on the Albireo ObsRO instrument from Weeks 0-4, Weeks 0-12, Weeks 0-22, Weeks 0-24, Weeks 0-36, Weeks 0-46, Weeks 0-48, Weeks 0-60, Weeks 0-70, or the proportion of positive pruritus assessments at each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 to Visit 12/Week 76 will be summarised descriptively as for the primary analysis for the US. Similar summaries will be provided based on AM scores as well as PM scores.

<sup>&</sup>lt;sup>7</sup> https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas.htm following CDC's method

<sup>8</sup> https://www.cdc.gov/nccdphp/dnpao/growthcharts/resources/sas-who.htm following WHO's method

<sup>&</sup>lt;sup>9</sup> Abdel-Rahman, Susan M et al. "Construction of Lambda, Mu, Sigma Values for Determining Mid-Upper Arm Circumference z Scores in U.S. Children Aged 2 Months Through 18 Years." Nutrition in clinical practice: official publication of the American Society for Parenteral and Enteral Nutrition vol. 32,1 (2017): 68-76.





The number and percent of patients achieving positive pruritus assessment for more than 50% of the time will be summarised by treatment group. Both AM and PM pruritus assessments will be included in the analysis of this endpoint. A cumulative distribution function (CDF) plot showing proportions of patients achieving positive pruritus assessment for more than X% of the time, X is the time of achieving positive pruritus assessment from 0 to 100%, by treatment group will be provided.

# Proportion of Responders for Pruritus Scores

The proportion of responders for pruritus scores will be tabulated by visit based on monthly scores and bi-weekly scores. The 95% CI of the proportion of responders will be provided, based on the exact method of Clopper-Pearson. A responder is defined as a patient who reports a decrease in pruritus score from unrounded baseline equivalent to or greater than the threshold of meaningful change estimated from the blinded psychometric analysis; the results of the blinded psychometric analysis across all anchors support a threshold of 1.0 point for AM, PM and AM and PM scratching scores. Baseline 1 and 2, defined in the table of derived variables in Appendix A, will be used for data analysis. Baseline 1 will only be used for patients in Cohort 1 who were on odevixibat in Study A4250-005.

# ❖ Biliary Diversion Surgery and Liver Transplantation

Number and percent of patients undergoing biliary diversion surgery and/or liver transplantation will be summarised by using descriptive statistics. A 95% CI also will be presented for the corresponding percentage. These parameters will be evaluated separately and together at Weeks 24, 48, 72 and all visits (every 16 weeks) during the optional extension period.

Kaplan-Meier curves will be used when appropriate for time-to-event data (that is, time to biliary diversion surgery or liver transplantation or death and time to any event). If a patient does not have any event, the patient will be censored at the last contact date. Median event-free times and associated 95% CIs will be calculated using Brookmeyer and Crowley methodology and a log-log transformation for constructing CIs.





#### ❖ Fibroscan<sup>®</sup>

The change in APRI and Fib-4 score will be summarised using descriptive statistics from baseline 2 to Week 72 and all visits (every 16 weeks) during the optional extension period.

#### ❖ PELD and MELD Score

The change in PELD and MELD will be summarised separately using descriptive statistics from baseline 2 to Week 72 and all visits (every 16 weeks) during the optional extension period.

#### UDCA and/or Rifampicin

Percentages of patients in use of UDCA and/or Rifampicin at weeks 24, 48, and 72 will be presented in 4 categories, use of UDCA, use of Rifampicin, use of UDCA or Rifampicin, use of UDCA and Rifampicin. Percentage will be based on patients in study at week 24, 48, and 72.

Shift tables from Baseline 2 in use of UDCA and/or Rifampicin at Weeks 24, 48, and 72 will be presented in the following categories. "None", "UCDA alone", "Rifampicin alone", "UCDA and Rifampicin", "Early Termination". Percentage will be based on patients in study at week 24, 48, and 72.

#### 9.6.5 Analyses of Exploratory Endpoints

The exploratory efficacy variables are listed in Section 4.3. All exploratory analyses mainly will be summarised descriptively based on the FAS, unless otherwise specified.

Exploratory variables including ALT; GGT; total bilirubin; INR; albumin; liver enzymes; leukocytes and platelets; measures of bile acid synthesis; Albireo PRO and ObsRO itching/scratching severity scores; Albireo PRO and ObsRO sleep parameters; Global Symptom Relief; and PedsQL will be summarised descriptively. For continuous data, the change from baseline will be analysed in addition to the presentation of actual visit values. For categorical data, shift tables or frequency and percentages of patients will be presented, as appropriate. A line graph of itching/scratching daily severity scores of Albireo PRO and ObsRO over time will be provided for each patient.





For continuous data, such as ALT; GGT; total bilirubin; INR; albumin; liver enzymes; leukocytes and platelets; measures of bile acid synthesis; and the total score and domain score of PedsQL, the change from baseline 2 will be analysed descriptively in addition to the actual visit values. Global Symptom Relief at Weeks 4, 12, 24, 48, 72 and all visits (every 16 weeks) during the optional extension period will be summarised as categorical variables. Time points (visit windows) are specified in Appendix B.

# Proportion of Positive Pruritus

The proportion of individual assessments meeting the definition of a positive pruritus assessment at the patient level on the Albireo PRO instrument completed by patients ≥8 years of age only will also be explored and summarised in a similar fashion as for the secondary endpoint, the proportion of individual assessments meeting the definition of a positive pruritus assessment at the patient level on the Albireo ObsRO instrument.

Change from baseline 2 in PRO/ObsRO itching and scratching severity scores will be summarised by each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76. A summary table will be provided for night-time scores and morning time scores separately.

The pooled pruritus score including observer-reported scratching for patients <8 years of age and patient-reported itch severity for patients  $\ge8$  years of age will be summarised in a similar manner.

The change from baseline 2 in PRO/ObsRO sleep parameters will be summarised at Week 72 as well as by each 4-week interval between Visit 1/Screening and Visit 5/Week 24, then by each visit between Visit 5/Week 24 and Visit 12/Week 76. Sleep parameters include difficulty of falling asleep and staying asleep, tiredness, and the number of awakenings.

#### ❖ Fibroscan<sup>®</sup>

Change from baseline 2 in stage of liver fibrosis measured by Fibroscan<sup>®</sup> will be analysed descriptively. The frequencies of stages will be summarised by shift tables. Steatosis grade analysis will be performed in a similar fashion. Liver fibrosis as assessed by post-treatment biopsy will be listed and change from baseline may be presented, if available.





#### Episodic Flares

Due to limited data availability and only 4 BRIC patients were enrolled in the study, the episodic flares data during the study will be presented as a listing.

# 9.7 Safety Analyses

All definitions relative to safety endpoints are detailed in Section 4.4.

All the safety analyses will be performed on the FAS for all safety variables specified below and summarised by cohort/treatment subgroup and overall.

For each safety variable, the last value collected before the first dose of study drug will be used as baseline (i.e., Baseline 2 defined in the table of derived variables in Appendix A) for all analyses unless otherwise specified.

In addition, different with efficacy analysis, laboratory related safety endpoints will be considered up to 28 days follow-up after the last dose.

#### 9.7.1 Adverse Events

All AEs will be classified by Primary SOC and PT according to MedDRA, Version 26.0 or higher.

AEs will be classified as TEAEs and defined as follows:

A TEAE is an AE occurring during the treatment period and within 28 days follow-up after the last dose that a) Has a start date on or after the first dose date of study drug, or b) Has a start date before the date of the first dose date of study drug, but worsened in severity on or after the date of the first dose date of study drug. If an AE started in Study A4250-005 and was ongoing at the time of enrolment in Study A4250-008, the AE will not be considered a TEAE unless it worsens in severity on or after the date of the first dose date of study drug.

AEs with missing start dates, but with stop dates that either overlap with the treatment period or are missing, will be considered TEAEs. A TEAE with missing drug relationship- will be considered as related. A TEAE with missing severity will be





considered as severe. Details for imputing missing or partial start dates of AEs are described in Appendix D.

For counting of the number of AEs, if 2 AE records have the same preferred term and the start date of the 2<sup>nd</sup> AE is the same as or next day after the end date of the 1<sup>st</sup> AE, then they will be counted as one AE only.

An overall summary of the incidence of TEAEs (number of patients with any events and number of events, if applicable) will include the following:

- All TEAEs
- Drug-related TEAEs (AE will be defined as drug-related if causality is either probably, possibly, or definitely related)
- Severe TEAEs
- TEAEs leading to study discontinuation
- Serious TEAEs
- Drug-related serious TEAEs
- TEAEs leading to death
- Any hepatic TEAEs
  - a. Any liver-related TEAE (events that, per the Investigator, are considered related to PFIC)
  - b. Any suspected drug-induced liver injury (DILI) TEAEs (as adjudicated by the Data Safety Monitoring Board [DSMB] and defined in Section 9.7.1.2)
  - c. Any TEAE of liver decompensation (as defined in Section 9.7.1.2)
  - d. Drug related hepatic disorders comprehensive search SMQ (narrow and broad)
- Any Fat-Soluble Vitamin Deficiency TEAEs refractory to clinically recommended vitamin supplementation (as defined in Section 9.7.1.1)
- Any Possible Sequelae of FSV Deficiency TEAEs by SOC and PT (Specified TEAEs with PTs are listed in Appendix G)





• Any Clinically Significant Diarrhoea TEAEs (as defined in Section 9.7.1.1)

TEAEs (number of patients with any events and number of events, if applicable) by SOC and PT in each treatment group will be tabulated for the following:

- TEAEs by SOC and PT including fat-soluble vitamin deficiencies, diarrhoea, hepatoxicity (as defined in Section 9.7.1.1). Note that hepatotoxicity will also be included with the tabulation of hepatic events
- All TEAEs by preferred term by descending incidence in Overall column
- TEAEs leading to study discontinuation by SOC and PT
- Serious TEAE by SOC and PT
- Drug-related serious TEAE by SOC and PT
- TEAEs leading to death by SOC and PT
- Common TEAEs (≥10% in overall)
- Hepatic TEAEs
  - a. Liver-related TEAEs (events that, per the Investigator, are considered related to PFIC) by SOC and preferred term
  - b. Suspected DILI events (as adjudicated by the DSMB and defined in Section 9.7.1.2)
  - c. TEAEs of liver decompensation (as defined in Section 9.7.1.2) by SOC and preferred term
  - d. Drug related hepatic disorders comprehensive search SMQ (narrow and broad)

Summary tables for the number of patients with any TEAEs by SOC and PT by severity (mild, moderate, severe) and by causality (related [possibly, probably and definitely] versus unrelated [unlikely and unrelated]), will also be provided during the treatment period. AEs with the worst severity will be used in the by-severity summaries. Similarly, AEs with the worst causality (related to treatment) will be used in the by-causality summaries. If severity or causality is missing, data will be imputed to the worst category.





Where a patient has the same AE, based on PT, reported multiple times in the treatment period, the patient will only be counted once at the PT level in AE frequency tables. Where a patient has multiple AEs within the same SOC in the treatment period, the patient will only be counted once at the SOC level in AE frequency tables.

In the AE summaries, AEs will be sorted alphabetically by SOC and PT. In addition, the numbers of patients with liver-related mortality, liver-decompensation events, and all-cause mortality will be presented using descriptive statistics. Kaplan-Meier curves may be used for time-to-event data (time taken to experience liver-decompensation event, all-cause mortality, and biliary diversion surgery in weeks).

All AEs (including pre-treatment and post-treatment AEs), serious adverse events (SAEs), and deaths will be listed. Separate listings for AEs leading to dose interruption, AEs listing to dose change, and AEs of Interest (Fat-Soluble Vitamin Deficiency, Diarrhoea, Hepatic AEs, and Possible Sequelae of Fat-Soluble Vitamin Deficiency as defined below) will also be provided.

# 9.7.1.1 Definition for TEAEs of Fat-Soluble Vitamin Deficiency, Diarrhoea, and Hepatotoxicity

The following TEAEs have been defined based on the population under study:

- New or worsening of fat-soluble vitamin deficiency refractory to clinically recommended vitamin supplementation.
  - All Investigator-reported verbatim terms related to decreases in vitamin levels or vitamin deficiency (e.g., preferred term of hypovitaminosis, Vitamin A decreased, Vitamin A deficiency) with the relevant concomitant medication records reviewed by the Medical Monitor, queried as needed, and the appropriate MedDRA preferred terms reported.
- Clinically significant diarrhoea, defined as any of the following:
  - Diarrhoea that persists for 21 or more days without any other aetiology based on medical review of other concurrent AEs for possible other causes of the diarrhoea or diagnostic testing (e.g., viral infections)





- Reported by the Investigator as severe in intensity or reported as an SAE due to the requirement for hospitalisation or as an important medical event
- Diarrhoea with concurrent dehydration requiring treatment with oral or intravenous rehydration and/or other treatment intervention based on medical review of AEs and concomitant medications
- Hepatoxicity: based on the SMQ of *Drug Related Hepatic Disorders*—comprehensive search SMQ (narrow and broad)
- Possible Sequelae of FSV Deficiency: based on the Specified TEAEs with PTs are listed in Appendix G.

For each of these categories, tabular summaries will be presented by MedDRA SOC and PT; the tables will also include the overall incidence of these AEs. Listings of patients with each of the events as defined will be provided.

# 9.7.1.2 Definitions and Determination of Hepatic Events

A DSMB was formed to independently assure the safety of patients enrolled in Study A4250-008, as well as to evaluate the integrity of study conduct and the data generated. The DSMB reviews the safety data at regular, pre-defined intervals and on an ad hoc basis as needed and makes recommendations regarding patient safety and study continuance (continuation, modification, or termination of the study). The DSMB is comprised of three paediatric hepatologists and an unblinded biostatistician.

As requested by the FDA, the DSMB has been chartered to review data from patients with hepatic AEs, including cases of suspected DILI and patients with liver decompensation events as defined below. The DSMB also reviews events that are reported in the SMQ of *Drug Related Hepatic Disorders; Severe Events Only*. The DSMB reviews each case and provides their expert opinion on the aetiology of the event.

For this review, Albireo prepares slides for presentation at the DSMB meeting on each patient who meets the criteria for hepatic event adjudication. Relevant liver-related laboratory values over time and a narrative summary of relevant information is provided to the DSMB. During the open session of the meeting, an Albireo physician reviews each case with the DSMB members, responds to questions, and/or obtains any additional





information requested by the DSMB. Albireo's assessment of the hepatotoxicity aetiology is documented for each event. During the closed session, the DSMB independently assesses the event aetiology which is documented on a Hepatic Event Adjudication Form that is attached to the meeting minutes. If the DSMB requests follow-up information, this is provided at the next scheduled meeting. The Adjudication Process Document outlines the events that will be adjudicated.

#### 9.7.1.2.1 Suspected Drug-Induced Liver Injury

As outlined in the protocol for Study A4250-008, patients with laboratory criteria that meet any of the following are considered suspected events of DILI and undergo review and adjudication of the event aetiology by the DSMB:

- ALT or AST ≥5 × ULN if ALT or AST was normal at Baseline, or an absolute threshold of 800 U/L, whichever comes first
- ALT or AST ≥3 × Baseline if ALT or AST was abnormal at Baseline, or an absolute threshold of 800 U/L, whichever comes first
- ALT or AST ≥3 × Baseline or an absolute threshold increases of +300 U/L, whichever comes first, and total bilirubin >2 × ULN if total bilirubin was normal at Baseline
- ALT or AST >5 × ULN if they are normal at Baseline, or absolute threshold increases of +300 U/L if ALT or AST > ULN at Baseline in presence of normal LDH and CPK
- Doubling of total bilirubin if total bilirubin was <3 mg/dL at Baseline and total bilirubin is greater than 2 × ULN unrelated to hemolysis or established genetic diseases, such as Gilbert's Syndrome.
- Increase in total bilirubin by >3 mg/dL if total bilirubin was  $\ge 3$  mg/dL at Baseline
- INR increase to >1.5 if INR was normal at Baseline and increase is refractory to Vitamin K administration
- INR increase by >0.4 if INR was abnormal at Baseline and increase is refractory to Vitamin K administration





 Any increase in total bilirubin and transaminases if accompanied by either a symptom of clinical hepatitis (vomiting, nausea, right upper quadrant pain) or immunological reaction (rash or 5% eosinophilia)

#### 9.7.1.2.2 Liver Decompensation Adverse Events

Events either identified by Investigators or meeting the Albireo definition of liver decompensation will undergo review and adjudication by the DSMB. Patients who meet either of the following criteria undergo review and adjudication of the event aetiology by the DSMB for liver decompensation:

- INR elevation >1.5 that is refractory to vitamin K administration
- In a patient with portal hypertension and cirrhosis, transition to decompensated cirrhosis evidenced by any of the following:
  - Presence of ascites
  - Hepatorenal syndrome
  - o Portopulmonary hypertension
  - Hepatopulmonary syndrome
  - Variceal haemorrhage
  - o Hepatic encephalopathy

#### 9.7.1.2.3 SMQ Drug-Related Hepatic Disorder AEs:

Events in the Standardised MedDRA query SMQ *Drug Related Hepatic Disorders; Severe Events Only* (SMQ No. 20000007) that are not captured in any of the above parameters will be presented to the DSMB for review.

The data of all adjudicated hepatic events provided by the DSMB will also be listed.





#### 9.7.2 Clinical Laboratory Evaluations

Clinical laboratory test results will be listed.

The following laboratory variables will be analyzed.

#### • Hematology:

- Red blood cells and platelets: hemoglobin, hematocrit, red blood cell count, and platelet count
- White blood cells: white blood cell count, neutrophils, lymphocytes, monocytes, basophils, and eosinophils

#### • Clinical chemistry:

- Metabolism: total cholesterol, triglycerides, creatine kinase, albumin
- Electrolytes: sodium, potassium, chloride, calcium
- Renal function: creatinine, blood urea nitrogen, estimated glomerular filtration rate
- Liver function: ALT, AST, Alkaline phosphatase (and isoenzymes as applicable), direct bilirubin, total bilirubin, gamma-glutamyl transferase
- Pregnancy test: Serum β-human chorionic gonadotropin (all female patients with positive urine pregnancy test)

#### Urinalysis:

- Urinalysis for quantitative analysis: pH, proteins, glucose, blood, ketones, leukocytes, and nitrites
- Other Labs: Vitamin A and E, 25-hydroxy vitamin D, INR, Alfa-fetoprotein (AFP), and Prothrombin Time

#### Quantitative Analyses

For all laboratory variables above, descriptive statistics for clinical laboratory values (in SI units for all tests, and in conventional units for selected tests (Appendix F) and absolute changes from baseline at each post-baseline visit (Appendix B) will be presented. The change to the last visit will also be summarized. Central laboratory data will be used for the summary. If central laboratory data are not available due to COVID-19 or other reasons, local laboratory data will be used, if available.

Change from baseline in ALT, AST, GGT, direct bilirubin, total bilirubin will be summarized by visit using descriptive statistics. Figure of mean (± standard error [SE])





changes from baseline 2 will be provided at each available post-baseline visit. The figures will only present results in a treatment group if there's data for at least 5 patients at that visit; if all treatment groups at that visit do not have at least 5 patients' data, that visit will not be presented in the figure.

Evaluation of drug-induced serious hepatotoxicity (eDISH) plots will be presented for baseline and post-baseline liver function (ALT vs total bilirubin). Baseline eDISH plot will present concurrent levels of baseline ALT vs. total bilirubin as multiples of upper limit of normal (ULN). Post-baseline eDISH plot will present concurrent levels of peak ALT on treatment vs. peak total bilirubin within 30 days of peak ALT as multiples of ULN. In addition, a modified eDISH plot will present concurrent peak ALT vs peak total bilirubin as multiples of individual patient baseline values. Corresponding summary tables will be provided.

Analyses according to reference normal range

Shift tables from baseline to the highest and lowest post-baseline value for quantitative variables will be presented for the clinical laboratory parameters. The laboratory results will be classified as low, normal, and high based on the normal range that was provided by central/local laboratories.

For ALT, AST and total bilirubin, a shift table based on the following classifications (per DILI guidance and CTCAE) will be presented:

• ALT and AST: ≤3 ULN, > 3 and ≤ 5 ULN, > 5 and ≤ 10 ULN, > 10 ULN Total Bilirubin: ≤2 ULN and > 2 ULN

#### Liver Monitoring

Furthermore, a listing of patients meeting the following criteria for liver monitoring will be provided as follows:

- (ALT or AST ≥3× baseline or absolute threshold increase ≥ 300 U/L) and total bilirubin >2 ULN (normal baseline) at the same visit
- ALT or AST >5 ULN (normal baseline) or increase ≥ 300 U/L (baseline ALT or AST > ULN) in presence of normal LDH and CPK at the same visit





- INR increased to >1.5 (normal baseline) or increased by >0.4 relative to baseline (abnormal baseline)
- Total bilirubin ≥2× baseline (baseline total bilirubin <3 mg/dL) and total bilirubin is greater than 2× ULN, or increased by ≥3 mg/dL relative to baseline (baseline total bilirubin ≥3 mg/dL)

### 9.7.3 Vital Sign Measurements

Descriptive statistics for vital signs (temperature, systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, weight, height/length, mid-arm circumference, and BMI) and changes from baseline in vital signs at each post-baseline visit will be presented in a summary table. The change to the last visit will also be summarised. A shift table for the number of patients with changes from baseline to the highest or lowest value (Appendix E) will be provided by cohort/treatment subgroup during the treatment period.

Vital signs data will be listed.

#### 9.7.4 Physical Examinations

All physical examination data (general appearance, eyes, ears, nose, throat, head/neck/thyroid, lymph nodes, cardiovascular, lungs/chest, abdomen, genitourinary, extremities, skin, musculoskeletal, neurological, and other body systems) will be summarised at each visit with percentages and frequencies along with abnormalities by cohort/treatment subgroup.

Abdominal ultrasound assessments for the liver, including Riedel's lobe, the portal vein, and the spleen also will be summarised descriptively for each visit.

Skin assessments on a 5-point scale (0-4 from no evidence of scratching to cutaneous bleeding, haemorrhage, scabbing) for face, right arm, left arm, right leg, left leg, and torso will be summarised at each visit with percentages and frequencies by cohort/treatment subgroup.

Physical examination and skin assessment data will be listed (including pre-treatment and post-treatment results).





#### 9.8 Other Analyses

# 9.8.1 Subgroup Analyses

Subgroup analyses will be performed for the primary efficacy endpoints for each of the following subgroups: age groups (<6 months, 6 months to 5 years, 6 to 12 years, and 13 to 18 years, >18 years), each PFIC type (1, 2, other, BRIC), region (US, EU, and RoW), sex, race, ethnicity, baseline serum bile acid (≥250 and <250 µmol/L), Child-Pugh classification, Bile Salt Export Pump (BSEP) type of PFIC 2 patients, and the use of UDCA, rifampicin (alone or either one). Subgroup analyses may be conducted for hepatic impairment classification per NCI Organ Dysfunction Working Group (ODWG) if appropriate.

# 9.8.2 Data Safety Monitoring Board

The DSMB will receive data in the form of tables, figures, and listings (provided by unblinded DSMB statistician from Firma who is independent to the Firma study team). The requirement for blinded or unblinded data is defined in the DSMB charter. Data provided to the DSMB will include, but is not limited to, demographics, baseline characteristics, medical and surgical history, prior and concomitant medications, AE and SAE data (by SOC and PT and by maximum intensity), laboratory data, liver monitoring, vital sign measurements, and abdominal ultrasound and patient disposition data.

#### 10. Changes to Planned Analysis from Study Protocol

The changes to the planned analysis in the protocol are listed below.

- 1. Endpoints
  - a. Removed below secondary efficacy endpoints
    - i. All-cause mortality
    - ii. Change in use of antipruritic medication at Weeks 24, 48, and 72
  - b. Added below secondary efficacy endpoints
    - i. Change in use of UDCA and/or Rifampicin at Weeks 24, 48, and 72
    - ii. Proportion of responders for pruritus scores





- c. Added below exploratory endpoint
  - Change from baseline in episodic flares during the study treatment for BRIC patients.
- d. Added below safety endpoint
  - i. All-cause mortality
- e. Updated secondary and exploratory efficacy endpoints to add the visits during extension period

# 2. Data Analysis

- a. For the number of patients with events (biliary diversion surgery or liver transplantation or death) and time to event, the comparison to the NAPPED population will be not included in this SAP and will be performed separately.
- b. The following analysis in the protocol "As an exploratory analysis of pruritus and serum bile acids, a comparison of treatment with A4250 120 μg/kg/day during the first 24 weeks of Study A4250-008 versus placebo patients over the 24week treatment period from Study A4250-005 will be carried out." was conducted in A4250 ISE analysis because Study A4250-008 did not have post-baseline data of Study A4250-005.
- 3. TEAE definition is updated from "during treatment period" to "during treatment period and within 28 days follow-up after the last dose".
- 4. Laboratory data will only be considered up to 14 days follow-up after the last dose of Odevixibat for efficacy related endpoints.
- **5.** For any hepatic TEAEs, add "Drug related hepatic disorders comprehensive search SMQ (narrow and broad)".





# 11. Appendices

# Appendix A: Derived Variables

A list of derived variables for demographic and baseline characteristics, various duration derivations, drug compliance, baseline derivations, and other important derivations applicable for this study is presented in Table 3.

Table 3: Derived Variables for Demographic and Baseline Characteristics, Various Duration Derivations, Drug Compliance, Baseline Derivations, and Other Important Derivations

| - | |
|---|---|
| VARIABLES | FORMULA |
| Demographic and Baseline Characteristics | |
| Age at informed consent (in years) | Cohort 1: For patients not from France and Germany, age will be calculated based on date of birth. For patients from France and Germany, only birth year was collected, and July 1 was imputed in the eDC system. The CRF collected age months and age years are based on the imputed date of birth. For analysis purpose, age will be calculated based on collected age months and age years on the Study A4250-005 CRF or the external file (primary source). Cohort 2: For patients not from France and Germany, age will be calculated based on date of birth. For patients from France and Germany, only birth year was collected, and July 1 was imputed in the eDC system. The CRF collected age months and age years are based on the imputed date of birth. For analysis purpose, age will be calculated based on collected age months and age years on the Study A4250-008 CRF or the external file (primary source). |
| BMI (kg/m²) | Weight (kg)/[height (m²) |
| PFIC diagnosis (in years) | Will be derived by SAS YRDIF function YRDIF (date of diagnosis of PFIC, date of informed consent, 'ACT/ACT') |
| Derivation of Duration | |
| Study day at any visit | Date of interest-date of first dose of study drug. One day is added if this difference is $\geq 0$ |
| Extent of exposure (days) | Date of last study drug intake-date of first study drug intake + 1 |
| Drug Compliance | |
| Compliance based on<br>CRF data | $100 \times [(total\ number\ of\ capsules\ dispensed-total\ number\ of\ capsules\ returned)\ /(total\ number\ of\ capsules\ planned\ to\ be\ taken)].$ This will be considered as the primary compliance rate. |
| Compliance based on<br>eDiary data up to week<br>24 | $100 \times$ (total number of capsules taken up to week 24/total number of capsules planned to be taken up to week 24). |





| VARIABLES | FORMULA |
|---|---|
| | The number of capsules planned to be taken will be estimated based on patient's body weight per Protocol Table 3. If a patient's weight changes at any time during the study, dose adjustment will be required. |
| Derivations for Efficacy | Parameters |
| Baseline (general) | Baseline 1 is defined as the last value prior to the first dose in Study A4250-005 for patients in Cohort 1. |
| | Baseline 2 is defined as the last value prior to the first dose in Study A4250-008 for all patients. For patients in Cohort 1, the pre-dose assessments of Study A4250-008 can be from Study A4250-005. |
| | Baseline 2 will be used in all analyses unless otherwise specified. |
| Baseline for serum bile<br>acids change from<br>baseline | Baseline 1 is defined for patients in Cohort 1 and will be calculated as the average of last 2 values prior to the first dose in Study A4250-005. If only one non-missing value is available, it will be used as baseline. |
| | Baseline 2 is defined as follows: Cohort 1: the average of the last 2 values before the first dose of study drug in Study A4250-008. In general, these 2 values are the values of the last 2 assessments of Study A4250-005. If pre-dose assessments are collected in Study A4250-008 for a patient, then the values of pre-dose assessments in Study A4250-008 will be considered first and used to calculate the baseline. These 2 values need to be taken from 2 consecutive scheduled visits or unscheduled visits. If only one value is available from 2 consecutive scheduled visits or unscheduled visits, then that value will be used as baseline. Cohort 2: the average of last 2 values prior to the first dose in Study A4250-008. If only one non-missing value is available, it will be used as baseline. Baseline 2 will be used in all analyses unless otherwise specified. |
| End value for serum bile<br>acids change from<br>baseline | The end value is the average of the values at Weeks 70 and 72 after the start of treatment. (Appendix B). If one value is missing, then the non-missing value will be used as the end value. If both values are missing, then the end value is missing. |
| Baseline, daily, weekly,<br>and monthly score by<br>AM and PM respectively<br>(scratching, itch<br>severity) | For both the Albireo ObsRO scratching item and the Albireo PRO itch severity score: All non-missing AM scores from the period of 14 days before or on the first dose day of study medications will be averaged as baseline. All non-missing PM scores from the period of 14 days before the first dose day of study medications will be averaged as baseline. Baseline score will be considered missing if ≥8 out of 14 assessments in the 14 days are missing (i.e. 50% rule is applied based on the number of planned assessments). A weekly AM (PM) score will be calculated by averaging all non-missing AM (PM) scores in a week. A weekly score will be considered missing if ≥4 out of 7 AM (PM) scores in a week are missing. |





| *** | <b>7</b> |
|---|---|
| VARIABLES | FORMULA |
| | A monthly AM (PM) score will be calculated by averaging all non-missing AM (PM) scores in a month (28 days). A monthly score will be considered missing if ≥15 out of 28 AM (PM) scores a week are missing. |
| | An AM (PM) average score at each visit after Week 24 will be calculated by averaging all non-missing AM (PM) scores between 2 visits with analysis windows applied (Appendix B). 50% rule is applied based on the number of planned assessments. |
| AM & PM baseline,<br>daily, weekly, and | For both the Albireo ObsRO scratching item and the Albireo PRO itch severity score: |
| monthly score<br>(scratching, itch | A daily AM & PM score will be averaged from the 2 ratings for each day. A daily score will be considered missing if both assessments are missing. |
| severity) | A weekly score will be calculated by averaging all non-missing AM and PM scores in a week. A weekly score will be considered missing if ≥8 out of 14 assessments in a week are missing. |
| | A monthly score will be calculated by averaging all non-missing AM and PM scores in a month (28 days). A monthly score will be considered missing if ≥29 out of 56 assessments in a month are missing. |
| | An average score of AM & PM at each visit after Week 24 will be calculated by averaging all non-missing AM and PM scores between 2 visits with analysis windows applied (Appendix B). 50% rule is applied based on the number of planned assessments. |
| | All non-missing AM scores from the period of 14 days before or on the first dose day of study medications, and all non-missing PM scores from the period of 14 days before the first dose day of study medications will be averaged as the AM & PM baseline score. Baseline score will be considered missing if ≥15 out of 28 assessments in the 14 days are missing. Rounded baseline score will be used for the analysis. |
| | One thing of note: |
| | Inclusion criteria No. 4 in Study A4250-005: |
| | Cohort 1: Patient must have history of significant pruritus and a caregiver-reported observed scratching in the eDiary average of ≥2 (on 0 to 4 scale) in the 2 weeks prior to randomisation in Study A4250-005. |
| | Inclusion criteria No. 4 in Study A4250-008: |
| | Cohort 2: Patient must have history of significant pruritus and a caregiver-reported observed scratching or patient reported itching (for patients >18 with no caregiver-reported observed scratching) in the eDiary average of $\geq$ 2 (on 0 to 4 scale) in the 2 weeks prior to the screening/inclusion visit (Visit 1) in Study A4250-008. |
| | The pruritus score for purposes of establishing eligibility was calculated by taking the average of the worse of the two scores for each day. The values for week one were averaged and the values for week 2 were averaged. The two weekly averages were then averaged to provide a single score. If this score was ≥2 the pruritus eligibility requirement was met. The calculation of pruritus eligibility score is different from the calculation of the baseline pruritus score defined in the SAP. |





| VARIABLES | FORMULA |
|---|---|
| Average of change from<br>baseline from each AM<br>and PM scores<br>(scratching, itch | The calculation below is based on the change from baseline in each AM and PM score. The values based on this calculation will be used for data analysis. |
| severity) | Change from baseline (daily) will be calculated by averaging all non-<br>missing values of change from baseline (AM and PM) in a day. A daily<br>change from baseline will be considered missing if both AM and PM<br>change from baseline in a day are missing. |
| | Change from baseline (weekly) will be calculated by averaging all non-missing values of change from baseline (AM and PM) in a week. A weekly change from baseline will be considered missing if ≥8 out of 14 change from baseline values in a week are missing. |
| | Change from baseline (monthly) will be calculated by averaging all non-missing values of change from baseline (AM and PM) in a month (28 days). A monthly change from baseline will be considered missing if ≥29 out of 56 assessments in a month are missing. |
| | Change from baseline at each visit after Week 24 will be calculated by averaging all non-missing values of change from baseline (AM and PM) between 2 visits with analysis windows applied (Appendix B). 50% rule is applied based on the number of planned assessments. |
| Baseline, daily, weekly,<br>and monthly (sleep<br>parameters, such as<br>difficulty falling asleep<br>and staying asleep,<br>tiredness, the number of<br>awakenings) | For patient- and observer-reported outcome scores of sleep parameters, the same approach above will be used as for scratching/itch severity by AM and PM, respectively, since there is just one rating per day. |
| Proportion of positive pruritus assessments | No imputation will be made for any missing data. The assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) will be treated as missing and excluded from analysis. The proportion of positive pruritus assessments will be calculated based on reported eDiary data only. 50% rule will be applied based on the number of planned assessments (Appendix B). |





| VARIABLES | FORMULA |
|---|---|
| Baseline for proportion of responders for | Baseline 1 is defined as the average of all non-missing daily scores from 14 days prior to the first dose of study drug in study A4250-005. |
| pruritus scores | Baseline 2 is defined as the average of all non-missing daily scores from 14 days prior to the first dose of study drug in study A4250-008 (For patients in Cohort 1, the pre-dose assessments of Study A4250-008 can be from Study A4250-005). |
| | Baseline score will be considered missing if $\geq 8$ out of 14 assessments in the 14 days are missing. The unrounded baseline score will be used for the analysis. |
| Derivations for Safety Pa | <br>arameters |
| AE duration (days) | AE end date-AE start date + 1 |
| TEAEs | An AE (classified by preferred term) occurring during the treatment period and within 28 days follow-up after the last dose that a) has a start date on or after the first dose date of study drug, or b) has a start date before the date of the first dose date of study drug, but worsened in severity on or after the date of the first dose date of study drug. If an AE started in Study A4250-005 and was ongoing at the time of enrolment in Study A4250-008, the AE will not be considered a TEAE unless it worsens in severity on or after the date of the first dose date of study drug. |

AE: adverse event; BMI: body mass index; CRF: case report form; eDiary: electronic diary; ObsRO: observer-reported outcome; PFIC: progressive familial intrahepatic cholestasis; PRO: patient-reported outcome; SAP: statistical analysis plan; TEAEs: treatment-emergent adverse events





# Appendix B: Visit Window

The observation closest to the target day is the measurement used in the analysis for each visit. The following visit window will apply for all laboratory parameters, questionnaires, vital signs, physical measurements and other efficacy parameters in the study, if not otherwise specified.

Table 4: Analysis Visit Window (General)

| TIMING OF ASSESSMENT (DAYS RELATIVE TO TREATMENT) | VISIT NAME TO<br>DISPLAY FOR<br>ANALYSIS | TARGET<br>DAY | STUDY DAY<br>(RELATIVE DAY) |
|---|---|---|---|
| Screening (Days -56 to -1) | Baseline | | ≤-1 |
| Day 1 Week 1 | Baseline | | 1 (Pre-dose) |
| Week 4 (± 5 days) | Week 4 | 28 | Post-baseline - 56 |
| Week 12 (± 7 days) | Week 12 | 84 | 57–119 |
| Week 22 (± 7 days) | Week 22 | 154 | 120–161 |
| Week 24 (± 7 days) | Week 24 | 168 | 162–210 |
| Week 36 (± 7 days) | Week 36 | 252 | 211–287 |
| Week 46 (± 7 days) | Week 46 | 322 | 288–329 |
| Week 48 (± 7 days) | Week 48 | 336 | 330–378 |
| Week 60 (± 7 days) | Week 60 | 420 | 379–455 |
| Week 70 (± 7 days) | Week 70 | 490 | 456–497 |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 498–(Last dose day + 14) |
| 4 weeks post last dose of study drug<br>(±7 days) | Follow-up | 28 post last<br>dose | Last dose day + 15—Last<br>dose day + 28 |
| For patients who enter optional extension period: | | | |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 498– Min(518, start day<br>of optional extension<br>period -1) |
| Week 88 | Week 88 | 616 | Min(519, start day of<br>optional extension<br>period)–672 |
| Week 104, 120, (continue every 16 weeks) | Week 104, 120,<br>(continue every 16<br>weeks) | 7*week # | (7*(week # - 8) + 1) –<br>Min(7*(week # + 8), Last<br>dose day + 14) |





Table 5: Analysis Visit Windows for GIC/GIS, Physical Measurements and Selected Lab Test)

| TIMING OF ASSESSMENT (DAYS RELATIVE TO TREATMENT) | VISIT NAME TO<br>DISPLAY FOR<br>ANALYSIS | TARGET<br>DAY | STUDY DAY<br>(RELATIVE DAY) |
|---|---|---|---|
| Screening (Days -56 to -1) | Baseline | | ≤-1 |
| Day 1 Week 1 | Baseline | | 1 (Pre-dose) |
| Week 4 (± 5 days) | Week 4 | 28 | Post-baseline - 56 |
| Week 12 (± 7 days) | Week 12 | 84 | 57–126 |
| Week 24 (± 7 days) | Week 24 | 168 | 127–252 |
| Week 48 (± 7 days) | Week 48 | 336 | 253-420 |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 421–(Last dose day + 14) |
| 4 weeks post last dose of study drug<br>(±7 days) | Follow-up | 28 post last<br>dose | Last dose day + 15-Last<br>dose day + 28 |
| For patients who enter optional exte | ension period: | | |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 421- Min(518, start day<br>of optional extension<br>period -1) |
| Week 88 | Week 88 | 616 | Min(519, start day of<br>optional extension<br>period)–672 |
| Week 104, 120, (continue every 16 weeks) | Week 104, 120,<br>(continue every 16<br>weeks) | 7*week# | (7*(week # - 8) + 1) –<br>Min(7*(week # + 8), Last<br>dose day + 14) |

Note: Physical measurements include physical examination, voluntary photography and skin examination. Selected lab tests include urinalysis and autotaxin, p-C4.





Table 6: Analysis Visit Window for PedsQL, Fibroscan, Abdominal Ultrasound and AFP

| TIMING OF ASSESSMENT (DAYS RELATIVE TO TREATMENT) | VISIT NAME TO<br>DISPLAY FOR<br>ANALYSIS | TARGET<br>DAY | STUDY DAY<br>(RELATIVE DAY) |
|---|---|---|---|
| Screening (Days -56 to -1) | Baseline | | ≤-1 |
| Day 1 Week 1 | Baseline | | 1 (Pre-dose) |
| Week 24 (± 7 days) | Week 24 | 168 | 71 –252 |
| Week 48 (± 7 days) | Week 48 | 336 | 253-420 |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 421–(last dose day + 14) |
| 4 weeks post last dose of study drug<br>(±7 days) | Follow-up | 28 post last<br>dose | Last dose day + 15—Last<br>dose day + 28 |
| For patients who enter optional exte | nsion period: | | |
| Week 72/EOT (± 7 days) | Week 72 | 504 | 421- Min(518, start day<br>of optional extension<br>period -1) |
| Week 88 | Week 88 | 616 | Min(519, start day of<br>optional extension<br>period)–672 |
| Week 104, 120, (continue every 16 weeks) | Week 104, 120,<br>(continue every 16<br>weeks) | 7*week # | (7*(week # - 8) + 1) –<br>Min(7*(week # + 8), Last<br>dose day + 14) |

For laboratory and non-laboratory parameters, if a patient has more than one measurement included within a window, the assessment closest to the target day will be used. In case of ties between observations located on different sides of the target day, the earlier assessment will be used. For laboratory parameters, central laboratory results will be used over local laboratory results if both are in a same analysis window.

Derivations for pruritus and other itching, scratching, sleep parameters measured by Albireo ObsRO and PRO instruments will be derived based on the following analysis window. For analysis purposes, diary entries will be assigned to a study day based on the recorded date regardless of recorded time. Please refer to the derivations in the table of derived variables in Appendix A for details.





Table 7: Analysis Visit Window for eDiary Parameters

| 4-WEEK/BY-VISIT<br>INTERVAL | INTERVALS TO INCLUDE<br>EDIARY DATA (DAYS) <sup>a</sup> | INTERVALS WITH >=50% OF EXPECTED DATA TO INCLUDE PATIENTS <sup>b</sup> (# OF EXPECTED DAYS TO REPORT EDIARY) |
|---|---|---|
| Weeks 1-4 | 1 - 28 | Weeks 1 – 4 (28 days) |
| Weeks 5 – 8 | 29 – 56 | Weeks 5 – 8 (28 days) |
| Weeks 9 – 12 | 57 – 84 | Weeks 9 – 12 (28 days) |
| Weeks 13 – 16 | 85 – 112 | Weeks 13 – 16 (28 days) |
| Weeks 17 – 20 | 113 – 140 | Weeks 17 – 20 (28 days) |
| Weeks 21 – 24 | 141 – 168 | Weeks 21 – 24 (28 days) |
| Weeks 34 – 36 | 169 – 287 | Weeks 31 – 41 (21 days) |
| Weeks 44 – 46 | 288 – 322 | Weeks 42 – 46 (21 days) |
| Weeks 47 – 48 | 323 – 378 | Weeks 47 – 54 (14 days) |
| Weeks 58 – 60 | 379 – 455 | Weeks 55 – 65 (21 days) |
| Weeks 68 - 70 | 456 – 490 | Weeks 66 – 70 (21 days) |
| Weeks 71 – 72 | 491 – 504 | Weeks 71 – 72 (14 days) |
| Weeks 72 – 76 | >=505 | >=505 (28 days) |

<sup>&</sup>lt;sup>a</sup> The proportion of positive pruritus assessments is calculated based on reported data only. The assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) will be excluded from the calculation.

<sup>&</sup>lt;sup>b</sup> To have an appropriate analysis, only include patients who reported at least 50% of expected data during the interval. Of notes, for Weeks 34-36, while eDiary data during weeks 25 to 41 will be included for analysis, 50% rule is applied to Weeks 31-41 only to make sure that a patient is on treatment long enough for the analysis of Weeks 34-36.





Table 8: Analysis Visit Window for Proportion of Responders for Pruritus Monthly Scores

| 4-WEEK/BY-VISIT<br>INTERVAL | INTERVALS TO INCLUDE<br>EDIARY DATA (DAYS) <sup>a</sup> | INTERVALS WITH >=50% OF<br>EXPECTED DATA TO INCLUDE<br>PATIENTS <sup>b</sup> (# OF EXPECTED<br>DAYS TO REPORT EDIARY) |
|---|---|---|
| Weeks 1-4 | 1 - 28 | Weeks 1 – 4 (28 days) |
| Weeks 5 – 8 | 29 – 56 | Weeks 5 – 8 (28 days) |
| Weeks 9 – 12 | 57 – 84 | Weeks 9 – 12 (28 days) |
| Weeks 13 – 16 | 85-112 | Weeks 13 – 16 (28 days) |
| Weeks 17 – 20 | 113 – 140 | Weeks 17 – 20 (28 days) |
| Weeks 21 – 24 | 141 – 168 | Weeks 21 – 24 (28 days) |
| Weeks 34 – 36 | 169 – 287 | Weeks 31 – 41 (21 days) |
| Weeks 45 – 48 | 288 - 378 | Weeks 42 – 54 (28 days) |
| Weeks 58 - 60 | 379 – 455 | Weeks 55 – 65 (21 days) |
| Weeks 68 – 72 | 456 – 504 | Weeks 66 – 72 (28 days) |

<sup>&</sup>lt;sup>a</sup> The proportion of responders for pruritus monthly scores is calculated based on reported data only. The assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) will be excluded from the calculation. <sup>b</sup> To have an appropriate analysis, only include patients who reported at least 50% of expected data during the interval. Of notes, for Weeks 34 − 36, while eDiary data during weeks 25 to 41 will be included for analysis, 50% rule is applied to Weeks 31 − 41 only to make sure that a patient is on treatment long enough for the analysis of Weeks 34 − 36.

Table 9: Analysis Visit Window for Proportion of Responders for Pruritus Biweekly Scores

| BI-WEEKLY/BY-VISIT<br>INTERVAL | INTERVALS TO INCLUDE<br>EDIARY DATA (DAYS) <sup>a</sup> | INTERVALS WITH >=50% OF<br>EXPECTED DATA TO INCLUDE<br>PATIENTS <sup>b</sup> (# OF EXPECTED<br>DAYS TO REPORT EDIARY) |
|---|---|---|
| Weeks 1 – 2 | 1 - 14 | Weeks 1 – 2 (14 days) |
| Weeks 3 – 4 | 15 - 28 | Weeks 3 – 4 (14 days) |
| Weeks 5 – 6 | 29 – 42 | Weeks 5 – 6 (14 days) |
| Weeks 7 – 8 | 43 – 56 | Weeks 7 – 8 (14 days) |
| Weeks 9 – 10 | 57 – 70 | Weeks 9 – 10 (14 days) |
| Weeks 11 – 12 | 71 – 84 | Weeks 11 – 12 (14 days) |
| Weeks 13 – 14 | 85 – 98 | Weeks 13 – 14 (14 days) |
| Weeks 15 – 16 | 99 – 112 | Weeks 15 – 16 (14 days) |
| Weeks 17 – 18 | 113 – 126 | Weeks 17 – 18 (14 days) |
| Weeks 19 – 20 | 127 – 140 | Weeks 19 – 20 (14 days) |
| Weeks 21 – 22 | 141 – 154 | Weeks 21 – 22 (14 days) |
| Weeks 23 – 24 | 155 – 168 | Weeks 23 – 24 (14 days) |
| Weeks 35 – 36 | 239 - 252 | Weeks 35 – 36 (14 days) |
| Weeks 47 – 48 | 323 – 336 | Weeks 47 – 48 (14 days) |
| Weeks 59 – 60 | 407 – 420 | Weeks 59 – 60 (14 days) |
| Weeks 71 – 72 | 491 – 504 | Weeks 71 – 72 (14 days) |





Version v2.1; Date: 04Apr2024


<sup>a</sup> The proportion of responders for pruritus bi-weekly scores is calculated based on reported data only. The assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) will be excluded from the calculation. <sup>b</sup> To have an appropriate analysis, only include patients who reported at least 50% of expected data during the interval. Of notes, for Weeks 35 − 36, while eDiary data during weeks 35 to 36 will be included for analysis, 50% rule is applied to Weeks 35 − 46 only to make sure that a patient is on treatment long enough for the analysis of Weeks 35 − 36.

Table 10: Analysis Visit Window for Proportion of Positive Pruritus Assessment

| CUMULATIVE<br>INTERVAL | INTERVALS TO INCLUDE<br>EDIARY DATA (DAYS) <sup>a</sup> (#<br>OF EXPECTED DAYS TO<br>REPORT EDIARY) | INTERVALS WITH >=50% OF<br>EXPECTED DATA TO INCLUDE<br>PATIENTS <sup>b</sup> (# OF EXPECTED<br>DAYS TO REPORT EDIARY) |
|---|---|---|
| Weeks 0 – 4 | 1 – 28 (28 days) | Weeks 1 – 4 (28 days) |
| Weeks 0 – 12 | 1 – 84 (84 days) | Weeks 9 – 12 (28 days) |
| Weeks 0 – 22 | 1 – 154 (154 days) | Weeks 19 – 22 (28 days) |
| Weeks 0 – 24 | 1 - 168 (168 days) | Weeks 21 – 24 (28 days) |
| Weeks 0 – 36 | 1 – 287 (189 days) | Weeks 31 – 41 (21 days) |
| Weeks 0 – 46 | 1 – 322 (210 days) | Weeks 42 – 46 (21 days) |
| Weeks 0 – 48 | 1 – 378 (224 days) | Weeks 47 – 54 (14 days) |
| Weeks 0 – 60 | 1 – 455 (245 days) | Weeks 55 – 65 (21 days) |
| Weeks 0 – 70 | 1 – 490 (266 days) | Weeks 66 – 70 (21 days) |
| Weeks 0 - 72 | 1 - 504 (280 days) | Weeks 71 – 72 (14 days) |

<sup>&</sup>lt;sup>a</sup> The proportion of positive pruritus assessments is calculated based on reported data only when >=50% of expected ediary data is reported. The assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) will be excluded from the calculation.

#### Appendix C: Definition of Region Variable

The list of country, country code, and region variable are provided in Table 11.

<sup>&</sup>lt;sup>b</sup> To have an appropriate analysis, only include patients who reported at least 50% of expected data during the interval. Of notes, for Weeks 0-36, while eDiary data during weeks 0 to 41 will be included for analysis, 50% rule is applied to Weeks 31-41 only to make sure than a patient is on treatment long enough for the analysis of Weeks 0-36.





Table 11: Definition of Region Variable

| COUNTRY | COUNTRY CODE | REGION VARIABLE |
|----------------|--------------|-----------------|
| Australia | AUS | RoW |
| Belgium | BEL | EU |
| Canada | CAN | RoW |
| France | FRA | EU |
| Germany | DEU | EU |
| Israel | ISR | RoW |
| Italy | ITA | EU |
| Netherlands | NLD | EU |
| Poland | POL | EU |
| Saudi Arabia | SAU | RoW |
| Spain | ESP | EU |
| Sweden | SWE | EU |
| Turkey | TUR | RoW |
| United Kingdom | GBR | EU |
| United States | USA | US |

EU: European Union; RoW: rest of world; US: United States

# Appendix D: Handling of Missing or Incomplete Dates

#### **Global Statement:**

If the imputed date is prior to the date of birth, then impute the missing date as date of birth.

Imputation rules for missing or partial AE start date are defined below:

# If only Day of AE start date is missing:

If the AE start year and month are the same as that for the first dose date, then:

• If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start day as the day of first dose date





• If AE end date is prior to first dose date, then impute the AE start day as 1

# If Day and Month of AE start date are missing:

If AE start year = first dose year, then:

- If the full (or partial) AE end date is NOT before the first dose date or AE end date is missing, then impute the AE start month and day as the month and day of first dose date
- If AE end date is prior to first dose date, then impute the AE start month as January and the day as 1

#### If Year of AE start date is missing:

If the year of AE start is missing or AE start date is completely missing, then query the site with no imputation. Also compare the full (or partial) AE end date to the first dose date. If the AE end date is before the first dose date, then the AE should be considered as a pre-treatment AE. Otherwise, the AE will be considered as TEAE.

Imputation rules for missing or partial non-study medication start/stop dates are defined below:

# Missing or partial non-study medication start date:

- If only day is missing, use the first day of the month
- If day and month are both missing, use the first day of the year
- If day, month, and year are all missing, use the date of the day before the first dose date

#### Missing or partial non-study medication stop date:

- If only day is missing, use the last day of the month
- If day and month are both missing, use the last day of the year
- If day, month, and year are all missing, assign "continuing" status to stop date





# Appendix E: Normal Reference Ranges of Vital Signs<sup>10</sup>

# Table 12: Heart Rate by Age (Beats/Minute) Reference

| AGE | AWAKE RATE |
|--------------------------|------------|
| Infant (<1 year) | 100-190 |
| Toddler (1-2 years) | 98-140 |
| Preschool (3-5 years) | 80-120 |
| School-age (6-11 years) | 75-118 |
| Adolescent (12-15 years) | 60-100 |
| > 15 years | 60-100 |

Table 13: Normal Respiratory Rate by Age (Breaths/Minute) Reference

| AGE | RESPIRATORY RATE |
|--------------------------|------------------|
| Infants (<1 year) | 30-53 |
| Toddler (1-2 years) | 22-37 |
| Preschool (3-5 years) | 20-28 |
| School-age (6-11 years) | 18-25 |
| Adolescent (12-15 years) | 12-20 |
| >15 years | 12-20 |

Table 14: Normal Blood Pressure by Age (mm Hg) Reference

| AGE | SYSTOLIC PRESSURE | DIASTOLIC PRESSURE |
|-----------------------------|-------------------|--------------------|
| Infant (<1 year) | 72-104 | 37-56 |
| Toddler (1-2 years) | 86-106 | 42-63 |
| Preschooler (3-5 years) | 89-112 | 46-72 |
| School-age (6-9 years) | 97-115 | 57-76 |
| Preadolescent (10-11 years) | 102-120 | 61-80 |
| Adolescent (12-15 years) | 110-131 | 64-83 |
| >15 years | 90-120 | 50-80 |

Statistical Analysis Plan Protocol A4250-008 Version v2.1; Date: 04Apr2024 

<sup>&</sup>lt;sup>10</sup> Pediatric Vital Signs Reference Chart. Peds cases - Pediatrics for Medical Students - Developed by Chris Novak and Peter Gill for PedsCases.com April 21, 2016 (http://www.pedscases.com/pediatric-vital-signsreference-Chart).





Table 15: Normal Temperature Range by Method

| МЕТНОВ | TEMPERATURE (°C) |
|----------------------------|------------------|
| Rectal | 36.6-38 |
| Ear | 35.8-38 |
| Oral | 35.5-37.5 |
| Axillary | 36.5-37.5 |
| Temporal/core <sup>a</sup> | 35.8-38 |

In the eCRF core and temporal temperature measurements can be ticked as methods. Rectal and Tympanic (ear) fall in this group. Additionally, temporal temperature measurements (using a temperature scanner on the forehead)—approximate closely to core temperature measurements and therefore can be classified in this category. For that reason, the normal temperature range for core and temporal temperature measurements will be defined as described.





# Appendix F: SI and US Conventional Units of Clinical Laboratory Values

| SERUM CHEMISTRY | SI UNIT | CONVENTIONAL UNIT |
|--------------------------|-------------|--------------------------|
| Analyte | · | |
| Alpha Fetoprotein | IU/mL | ng/mL |
| Direct bilirubin | μmol/L | mg/dL |
| Calcium | mmol/L | mg/dL |
| Chloride | mmol/L | mEq/L |
| Creatinine | μmol/L | mg/dL |
| Potassium | mmol/L | mEq/L |
| Sodium | mmol/L | mEq/L |
| Serum bile acid | μmol/L | μg/mL |
| Total bilirubin | μmol/L | mg/dL |
| Haematology | SI Unit | Conventional Unit |
| Analyte | | |
| Haematocrit | ratio (L/L) | % |
| Haemoglobin | g/L | g/dL |
| Red blood count (RBC) | x10^12/L | x10^6/μL |
| Platelet count | x10^9/L | x10^3/μL |
| White blood cell count | x10^9/L | x10^3/μL |
| Fat Soluble Vitamins | SI Unit | Conventional Unit |
| Vitamin A | μmol/L | ug/dL |
| Vitamin E | μmol/L | mg/L |
| Vitamin D (25-dihydroxy) | nmol/L | ng/mL |
| Vitamin K | nmol/L | ng/mL |
| Urinalysis | SI Unit | <b>Conventional Unit</b> |
| Analyte | | |
| Glucose | mmol/L | mg/dL |
| Ketones | mmol/L | mg/dL |
| Protein | mmol/L | mg/dL |




## Appendix G: PT Term of Possible Sequelae of FSV Deficiency

| PT Term | Code |
|--------------------------------------------------|----------|
| Acetabulum fracture | 10000397 |
| Activated partial thromboplastin time abnormal | 10000631 |
| Activated partial thromboplastin time prolonged | 10000636 |
| Adrenal haemorrhage | 10001361 |
| Alopecia | 10001760 |
| Anastomotic ulcer haemorrhage | 10002244 |
| Ankle fracture | 10002544 |
| Aortic aneurysm rupture | 10002886 |
| Areflexia | 10003084 |
| Arrhythmia | 10003119 |
| Arterial rupture | 10003173 |
| Auricular haematoma | 10003797 |
| Bleeding varicose vein | 10005144 |
| Blindness | 10005169 |
| Blindness transient | 10005184 |
| Blood blister | 10005372 |
| Blood calcium decreased | 10005395 |
| Blood urine | 10005863 |
| Bone pain | 10006002 |
| Brain stem haemorrhage | 10006145 |
| Breast haemorrhage | 10006254 |
| Broad ligament haematoma | 10006375 |
| Calcium deficiency | 10006956 |
| Cephalhaematoma | 10008014 |
| Cerebellar haemorrhage | 10008030 |
| Cerebral aneurysm ruptured syphilitic | 10008076 |
| Cerebral arteriovenous malformation haemorrhagic | 10008086 |
| Cerebral haemorrhage | 10008111 |
| Cerebral haemorrhage neonatal | 10008112 |
| Choroidal haemorrhage | 10008786 |
| Clavicle fracture | 10009245 |
| Closed fracture manipulation | 10009506 |
| Coagulation factor IX level decreased | 10009746 |
| Coagulation factor VII level decreased | 10009761 |
| Coagulation factor X level decreased | 10009775 |
| Coagulation time prolonged | 10009799 |





| PT Term | Code |
|----------------------------------------|----------|
| Coagulopathy | 10009802 |
| Colonic haematoma | 10009996 |
| Complicated fracture | 10010149 |
| Compression fracture | 10010214 |
| Congenital anomaly | 10010356 |
| Conjunctival haemorrhage | 10010719 |
| Corneal scar | 10011044 |
| Cystitis haemorrhagic | 10011793 |
| Decreased immune responsiveness | 10011968 |
| Dementia | 10012267 |
| Dental caries | 10012318 |
| Diarrhoea haemorrhagic | 10012741 |
| Disseminated intravascular coagulation | 10013442 |
| Diverticulitis intestinal haemorrhagic | 10013541 |
| Diverticulum intestinal haemorrhagic | 10013560 |
| Dry eye | 10013774 |
| Duodenal ulcer haemorrhage | 10013839 |
| Duodenitis haemorrhagic | 10013865 |
| Dwarfism | 10013883 |
| Dysarthria | 10013887 |
| Dysphagia | 10013950 |
| Ear haemorrhage | 10014009 |
| Ecchymosis | 10014080 |
| Encephalitis haemorrhagic | 10014589 |
| Enterocolitis haemorrhagic | 10014896 |
| Epistaxis | 10015090 |
| Exsanguination | 10015719 |
| External fixation of fracture | 10015741 |
| Extradural haematoma | 10015769 |
| Extravasation blood | 10015867 |
| Eye haemorrhage | 10015926 |
| Factor IX deficiency | 10016077 |
| Femoral neck fracture | 10016450 |
| Femur fracture | 10016454 |
| Fibula fracture | 10016667 |
| Foetal-maternal haemorrhage | 10016871 |
| Foot fracture | 10016970 |
| Forearm fracture | 10016997 |





| PT Term | Code |
|----------------------------------------|----------|
| Fracture | 10017076 |
| Fracture delayed union | 10017081 |
| Fracture malunion | 10017085 |
| Fracture nonunion | 10017088 |
| Fractured sacrum | 10017308 |
| Gait disturbance | 10017577 |
| Gastric haemorrhage | 10017788 |
| Gastric ulcer haemorrhage | 10017826 |
| Gastric ulcer haemorrhage, obstructive | 10017829 |
| Gastritis alcoholic haemorrhagic | 10017857 |
| Gastritis haemorrhagic | 10017866 |
| Gastrointestinal haemorrhage | 10017955 |
| Gingival bleeding | 10018276 |
| Greenstick fracture | 10018720 |
| Haemarthrosis | 10018829 |
| Haematemesis | 10018830 |
| Haematocoele | 10018833 |
| Haematochezia | 10018836 |
| Haematoma | 10018852 |
| Haematospermia | 10018866 |
| Haematuria | 10018867 |
| Blood urine present | 10018870 |
| Haematuria traumatic | 10018871 |
| Haemoperitoneum | 10018935 |
| Haemoptysis | 10018964 |
| Haemorrhage in pregnancy | 10018981 |
| Haemorrhage intracranial | 10018985 |
| Haemorrhage subcutaneous | 10018999 |
| Haemorrhage subepidermal | 10019001 |
| Haemorrhagic cerebral infarction | 10019005 |
| Haemorrhagic disease of newborn | 10019008 |
| Haemorrhagic disorder | 10019009 |
| Haemorrhagic infarction | 10019013 |
| Haemorrhagic stroke | 10019016 |
| Haemothorax | 10019027 |
| Hand fracture | 10019114 |
| Henoch-Schonlein purpura | 10019617 |
| Hepatic haematoma | 10019676 |





| PT Term | Code |
|------------------------------------------|----------|
| Hepatic haemorrhage | 10019677 |
| Hereditary haemorrhagic telangiectasia | 10019883 |
| Hip fracture | 10020100 |
| Humerus fracture | 10020462 |
| Hyphaema | 10020923 |
| Hypophosphataemia | 10021058 |
| Hyporeflexia | 10021089 |
| Ilium fracture | 10021343 |
| Impaired healing | 10021519 |
| Increased tendency to bruise | 10021688 |
| Injection site bruising | 10022052 |
| Injection site haematoma | 10022066 |
| Injection site haemorrhage | 10022067 |
| Intermenstrual bleeding | 10022559 |
| Internal fixation of fracture | 10022576 |
| International normalised ratio abnormal | 10022592 |
| International normalised ratio increased | 10022595 |
| Intracranial tumour haemorrhage | 10022775 |
| Intraventricular haemorrhage | 10022840 |
| Intraventricular haemorrhage neonatal | 10022841 |
| Keratomalacia | 10023361 |
| Kidney contusion | 10023413 |
| Kyphosis | 10023509 |
| Mallory-Weiss syndrome | 10026712 |
| Melaena | 10027141 |
| Menometrorrhagia | 10027295 |
| Mouth haemorrhage | 10028024 |
| Multiple fractures | 10028200 |
| Muscle haemorrhage | 10028309 |
| Muscle spasms | 10028334 |
| Muscular weakness | 10028372 |
| Musculoskeletal pain | 10028391 |
| Myalgia | 10028411 |
| Myocardial rupture | 10028604 |
| Nephritis haemorrhagic | 10029132 |
| Neuropathic arthropathy | 10029326 |
| Night blindness | 10029404 |
| Nipple exudate bloody | 10029418 |





| PT Term | Code |
|-----------------------------------|----------|
| Nystagmus | 10029864 |
| Oesophageal haemorrhage | 10030172 |
| Oesophageal ulcer haemorrhage | 10030202 |
| Oesophageal varices haemorrhage | 10030210 |
| Oesophagitis haemorrhagic | 10030219 |
| Open fracture | 10030527 |
| Open reduction of fracture | 10030682 |
| Open reduction of spinal fracture | 10030684 |
| Ophthalmoplegia | 10030875 |
| Optic disc haemorrhage | 10030919 |
| Optic nerve sheath haemorrhage | 10030941 |
| Orbital haemorrhage | 10031045 |
| Osteomalacia | 10031250 |
| Osteoporosis | 10031282 |
| Osteoporotic fracture | 10031290 |
| Ovarian haematoma | 10033263 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatitis haemorrhagic | 10033650 |
| Pathological fracture | 10034156 |
| Pelvic haematoma obstetric | 10034248 |
| Penile haemorrhage | 10034305 |
| Peptic ulcer haemorrhage | 10034344 |
| Pericardial haemorrhage | 10034476 |
| Perineal haematoma | 10034520 |
| Periorbital haematoma | 10034544 |
| Petechiae | 10034754 |
| Pharyngeal haemorrhage | 10034827 |
| Placenta praevia haemorrhage | 10035121 |
| Post abortion haemorrhage | 10036246 |
| Post-traumatic osteoporosis | 10036315 |
| Postpartum haemorrhage | 10036417 |
| Premature separation of placenta | 10036608 |
| Proctitis haemorrhagic | 10036778 |
| Prostatic haemorrhage | 10036960 |
| Prothrombin level abnormal | 10037048 |
| Prothrombin level decreased | 10037050 |
| Prothrombin time abnormal | 10037057 |
| Prothrombin time prolonged | 10037063 |





| PT Term | Code |
|----------------------------------------|----------|
| Pulmonary alveolar haemorrhage | 10037313 |
| Pulmonary contusion | 10037370 |
| Pulmonary haemorrhage | 10037394 |
| Purpura | 10037549 |
| Purpura fulminans | 10037556 |
| Purpura neonatal | 10037557 |
| Purpura senile | 10037560 |
| Radius fracture | 10037802 |
| Rectal haemorrhage | 10038063 |
| Rectal ulcer haemorrhage | 10038081 |
| Renal haematoma | 10038459 |
| Renal haemorrhage | 10038460 |
| Respiratory tract haemorrhage | 10038727 |
| Respiratory tract haemorrhage neonatal | 10038728 |
| Retinal haemorrhage | 10038867 |
| Retroperitoneal haemorrhage | 10038980 |
| Rib fracture | 10039117 |
| Ruptured cerebral aneurysm | 10039330 |
| Scrotal haematoma | 10039749 |
| Senile osteoporosis | 10039984 |
| Short stature | 10040600 |
| Spinal compression fracture | 10041541 |
| Spinal fracture | 10041569 |
| Splenic haematoma | 10041646 |
| Splenic haemorrhage | 10041647 |
| Splinter haemorrhages | 10041663 |
| Sternal fracture | 10042015 |
| Stomatitis haemorrhagic | 10042132 |
| Stress fracture | 10042212 |
| Subarachnoid haemorrhage | 10042316 |
| Subarachnoid haemorrhage neonatal | 10042317 |
| Subcutaneous haematoma | 10042345 |
| Subdural haematoma | 10042361 |
| Subdural haematoma evacuation | 10042363 |
| Subdural haemorrhage | 10042364 |
| Subdural haemorrhage neonatal | 10042365 |
| Third stage postpartum haemorrhage | 10043449 |
| Thrombocytopenic purpura | 10043561 |





| PT Term | Code |
|----------------------------------------------------|----------|
| Thrombotic thrombocytopenic purpura | 10043648 |
| Tibia fracture | 10043827 |
| Tongue haematoma | 10043959 |
| Tooth injury | 10044043 |
| Tooth malformation | 10044046 |
| Traumatic haematoma | 10044522 |
| Tremor | 10044565 |
| Ulna fracture | 10045375 |
| Umbilical haemorrhage | 10045455 |
| Upper gastrointestinal haemorrhage | 10046274 |
| Urinary bladder haemorrhage | 10046528 |
| Uterine haemorrhage | 10046788 |
| Vaginal haematoma | 10046909 |
| Vaginal haemorrhage | 10046910 |
| Varicose vein ruptured | 10046999 |
| Vascular purpura | 10047097 |
| Ventricle rupture | 10047279 |
| Vitamin A deficiency related conjunctival disorder | 10047588 |
| Vitamin A deficiency related corneal disorder | 10047589 |
| Vitreous haemorrhage | 10047655 |
| Vulval haematoma | 10047756 |
| Vulval haematoma evacuation | 10047757 |
| Withdrawal bleed | 10047998 |
| Wrist fracture | 10048049 |
| Xerophthalmia | 10048221 |
| Xerosis | 10048222 |
| Aneurysm ruptured | 10048380 |
| Atrial rupture | 10048761 |
| Myocardial haemorrhage | 10048849 |
| Nail bed bleeding | 10048891 |
| Spinal cord haemorrhage | 10048992 |
| Osteopenia | 10049088 |
| Fractured coccyx | 10049164 |
| Spinal epidural haemorrhage | 10049236 |
| Lip haemorrhage | 10049297 |
| Bone density decreased | 10049470 |
| Traumatic fracture | 10049514 |
| Anal haemorrhage | 10049555 |





| PT Term | Code |
|------------------------------------|----------|
| Urethral haemorrhage | 10049710 |
| Tumour haemorrhage | 10049750 |
| Pituitary haemorrhage | 10049760 |
| Shock haemorrhagic | 10049771 |
| Melaena neonatal | 10049777 |
| Tongue haemorrhage | 10049870 |
| Osteoporosis prophylaxis | 10049904 |
| Mediastinal haematoma | 10049941 |
| Cervical vertebral fracture | 10049946 |
| Lumbar vertebral fracture | 10049947 |
| Thoracic vertebral fracture | 10049948 |
| Cervix haematoma uterine | 10050020 |
| Cervix haemorrhage uterine | 10050022 |
| Urogenital haemorrhage | 10050058 |
| Application site bruise | 10050114 |
| Cerebral haemorrhage foetal | 10050157 |
| Spinal epidural haematoma | 10050162 |
| Spinal subdural haematoma | 10050164 |
| Application site purpura | 10050182 |
| Skin ulcer haemorrhage | 10050377 |
| Chronic gastrointestinal bleeding | 10050399 |
| Haematosalpinx | 10050468 |
| Scleral haemorrhage | 10050508 |
| Contusion | 10050584 |
| Lower gastrointestinal haemorrhage | 10050953 |
| Post procedural haemorrhage | 10051077 |
| Catheter site haemorrhage | 10051099 |
| Incision site haemorrhage | 10051100 |
| Puncture site haemorrhage | 10051101 |
| Parotid gland haemorrhage | 10051166 |
| Soft tissue haemorrhage | 10051297 |
| Carotid aneurysm rupture | 10051328 |
| Wound haemorrhage | 10051373 |
| Retinopathy haemorrhagic | 10051447 |
| Corneal bleeding | 10051558 |
| Haematoma infection | 10051564 |
| Testicular haemorrhage | 10051877 |
| Osteorrhagia | 10051937 |





| PT Term | Code |
|-----------------------------------------------------------------|----------|
| Urinary occult blood positive | 10052287 |
| Brain contusion | 10052346 |
| Large intestinal haemorrhage | 10052534 |
| Small intestinal haemorrhage | 10052535 |
| Meningorrhagia | 10052593 |
| Comminuted fracture | 10052614 |
| Induced abortion haemorrhage | 10052844 |
| Eyelid bleeding | 10053196 |
| Fracture displacement | 10053206 |
| Anticoagulant therapy | 10053468 |
| Traumatic haemorrhage | 10053476 |
| Vascular rupture | 10053649 |
| Growth retardation | 10053759 |
| Gastroduodenal haemorrhage | 10053768 |
| Cerebral haematoma | 10053942 |
| Vascular pseudoaneurysm ruptured | 10053949 |
| Epiphyseal fracture | 10053962 |
| Implant site haemorrhage | 10053995 |
| Vessel puncture site haemorrhage | 10054092 |
| Haemorrhagic tumour necrosis | 10054096 |
| Haemorrhoidal haemorrhage | 10054787 |
| Retroplacental haematoma | 10054798 |
| Hepatic haemangioma rupture | 10054885 |
| Pelvic haematoma | 10054974 |
| Pulmonary haematoma | 10054991 |
| Arteriovenous fistula site haemorrhage | 10055123 |
| Arteriovenous graft site haemorrhage | 10055126 |
| Arteriovenous fistula site haematoma | 10055150 |
| Arteriovenous graft site haematoma | 10055152 |
| Catheter site haematoma | 10055662 |
| Haemorrhagic transformation stroke | 10055677 |
| Haemorrhage | 10055798 |
| Haemorrhage coronary artery | 10055803 |
| Haemorrhage urinary tract | 10055847 |
| Postmenopausal haemorrhage | 10055870 |
| Haematoma muscle | 10055890 |
| Protein induced by vitamin K absence or antagonist II | 10056243 |
| Protein induced by vitamin K absence or antagonist II increased | 10056247 |





| PT Term | Code |
|----------------------------------------------|----------|
| Mediastinal haemorrhage | 10056343 |
| Anastomotic haemorrhage | 10056346 |
| Pituitary apoplexy | 10056447 |
| Intra-abdominal haematoma | 10056457 |
| Gastrointestinal ulcer haemorrhage | 10056743 |
| Body height decreased | 10056812 |
| Palpable purpura | 10056872 |
| Fracture debridement | 10057147 |
| Loss of proprioception | 10057332 |
| Ciliary body haemorrhage | 10057417 |
| Iris haemorrhage | 10057418 |
| Tonsillar haemorrhage | 10057450 |
| Ocular retrobulbar haemorrhage | 10057571 |
| Gastric varices haemorrhage | 10057572 |
| Fracture reduction | 10057609 |
| Cognitive disorder | 10057668 |
| Bloody discharge | 10057687 |
| Purpura non-thrombocytopenic | 10057739 |
| Peritoneal haematoma | 10058095 |
| Retroperitoneal haematoma | 10058360 |
| Spinal deformity | 10058907 |
| Thalamus haemorrhage | 10058939 |
| Putamen haemorrhage | 10058940 |
| Haemobilia | 10058947 |
| Acute haemorrhagic leukoencephalitis | 10058994 |
| Cullen's sign | 10059029 |
| Parathyroid haemorrhage | 10059051 |
| Papillary muscle haemorrhage | 10059164 |
| Intestinal haemorrhage | 10059175 |
| Haemorrhagic cyst | 10059189 |
| Adrenal haematoma | 10059194 |
| Infusion site bruising | 10059203 |
| Incision site haematoma | 10059241 |
| Intracranial haematoma | 10059491 |
| Haemorrhagic urticaria | 10059499 |
| Haemorrhagic ascites | 10059766 |
| Renal cyst haemorrhage | 10059846 |
| Anticoagulation drug level above therapeutic | 10060320 |





| PT Term | Code |
|---------------------------------------|----------|
| Skin neoplasm bleeding | 10060712 |
| Mesenteric haemorrhage | 10060717 |
| Haematoma evacuation | 10060733 |
| Haemorrhagic ovarian cyst | 10060781 |
| Aortic rupture | 10060874 |
| Arterial haemorrhage | 10060964 |
| Cerebellar haematoma | 10061038 |
| Pelvic fracture | 10061161 |
| Genital haemorrhage | 10061178 |
| Haemorrhage foetal | 10061191 |
| Intra-abdominal haemorrhage | 10061249 |
| Large intestinal ulcer haemorrhage | 10061262 |
| Mucosal haemorrhage | 10061298 |
| Pelvic deformity | 10061335 |
| Scrotal haemorrhage | 10061361 |
| Traumatic intracranial haemorrhage | 10061387 |
| Upper limb fracture | 10061394 |
| Vitamin A deficiency eye disorder | 10061412 |
| Scrotal haematocoele | 10061517 |
| Small intestinal ulcer haemorrhage | 10061550 |
| Ulcer haemorrhage | 10061577 |
| Lower limb fracture | 10061599 |
| Coagulation factor IX level abnormal | 10061770 |
| Coagulation factor VII level abnormal | 10061772 |
| Coagulation factor X level abnormal | 10061774 |
| Occult blood positive | 10061880 |
| Fracture treatment | 10061959 |
| Haemorrhage neonatal | 10061993 |
| Intracerebral haematoma evacuation | 10062025 |
| Knee deformity | 10062061 |
| Tracheal haemorrhage | 10062543 |
| Tooth fracture | 10062544 |
| Bladder tamponade | 10062656 |
| Haemorrhagic diathesis | 10062713 |
| Thoracic haemorrhage | 10062744 |
| Naevus haemorrhage | 10062955 |
| Haematotympanum | 10063013 |
| Post procedural haematoma | 10063188 |





| PT Term | Code |
|--------------------------------------------|----------|
| International normalised ratio fluctuation | 10063351 |
| Circulating anticoagulant positive | 10063576 |
| Graft haemorrhage | 10063577 |
| Catheter site bruise | 10063587 |
| Pelvic haemorrhage | 10063678 |
| Implant site haematoma | 10063780 |
| Vulval haemorrhage | 10063816 |
| Implant site bruising | 10063850 |
| Uterine haematoma | 10063875 |
| Vessel puncture site bruise | 10063881 |
| Anal ulcer haemorrhage | 10063896 |
| Polymenorrhagia | 10064050 |
| Angina bullosa haemorrhagica | 10064223 |
| Thyroid haemorrhage | 10064224 |
| Skin haemorrhage | 10064265 |
| Umbilical cord haemorrhage | 10064534 |
| Haemorrhagic arteriovenous malformation | 10064595 |
| Breast haematoma | 10064753 |
| Tooth socket haemorrhage | 10064946 |
| Eyelid haematoma | 10064976 |
| Ulcerative keratitis | 10064996 |
| Coital bleeding | 10065019 |
| Haemophilic arthropathy | 10065057 |
| Spontaneous haematoma | 10065304 |
| Venous haemorrhage | 10065441 |
| Infusion site haematoma | 10065463 |
| Infusion site haemorrhage | 10065464 |
| Bronchial haemorrhage | 10065739 |
| Laryngeal haemorrhage | 10065740 |
| Ovarian haemorrhage | 10065741 |
| Spermatic cord haemorrhage | 10065742 |
| Ureteric haemorrhage | 10065743 |
| Vessel puncture site haematoma | 10065902 |
| Torus fracture | 10066094 |
| Avulsion fracture | 10066184 |
| Post procedural haematuria | 10066225 |
| Bone contusion | 10066251 |
| Lip haematoma | 10066304 |





| PT Term | Code |
|-------------------------------------------------------|----------|
| Impacted fracture | 10066386 |
| Basal ganglia haemorrhage | 10067057 |
| Liver contusion | 10067266 |
| Cerebral microhaemorrhage | 10067277 |
| Astringent therapy | 10067372 |
| Abdominal wall haematoma | 10067383 |
| Haemostasis | 10067439 |
| Myelomalacia | 10067441 |
| Bloody peritoneal effluent | 10067442 |
| Decreased vibratory sense | 10067502 |
| Intrapartum haemorrhage | 10067703 |
| Haemorrhagic erosive gastritis | 10067786 |
| Abdominal wall haemorrhage | 10067788 |
| Haemorrhagic hepatic cyst | 10067796 |
| Gastric occult blood positive | 10067855 |
| Aortic intramural haematoma | 10067975 |
| Aortic dissection rupture | 10068119 |
| Pharyngeal haematoma | 10068121 |
| Application site haematoma | 10068317 |
| Choroidal haematoma | 10068642 |
| Splenic varices haemorrhage | 10068662 |
| Umbilical haematoma | 10068712 |
| Bone density abnormal | 10068789 |
| Anorectal varices haemorrhage | 10068925 |
| Periprosthetic fracture | 10069135 |
| Abnormal withdrawal bleeding | 10069195 |
| Vaccination site haematoma | 10069472 |
| Vaccination site haemorrhage | 10069475 |
| Vaccination site bruising | 10069484 |
| Subgaleal haematoma | 10069510 |
| Paranasal sinus haematoma | 10069702 |
| Loss of anatomical alignment after fracture reduction | 10069723 |
| Intestinal haematoma | 10069829 |
| Lacrimal haemorrhage | 10069930 |
| Penile haematoma | 10070656 |
| Muscle contusion | 10070757 |
| Atypical femur fracture | 10070884 |
| Laryngeal haematoma | 10070885 |





| PT Term | Code |
|----------------------------------------------------|----------|
| Subchorionic haemorrhage | 10071010 |
| Growth failure | 10071095 |
| Brain stem microhaemorrhage | 10071205 |
| Cerebellar microhaemorrhage | 10071206 |
| Procedural haemorrhage | 10071229 |
| Haemorrhagic vasculitis | 10071252 |
| Wound haematoma | 10071504 |
| Mesenteric haematoma | 10071557 |
| Post-traumatic punctate intraepidermal haemorrhage | 10071639 |
| Periorbital haemorrhage | 10071697 |
| Intraocular haematoma | 10071934 |
| Subretinal haematoma | 10071935 |
| Vitreous haematoma | 10071936 |
| Central nervous system haemorrhage | 10072043 |
| Fracture pain | 10072132 |
| Tooth pulp haemorrhage | 10072228 |
| Haemorrhagic thyroid cyst | 10072256 |
| Post transfusion purpura | 10072265 |
| Radiation associated haemorrhage | 10072281 |
| Atypical fracture | 10072395 |
| Subchorionic haematoma | 10072596 |
| Peripartum haemorrhage | 10072693 |
| Application site haemorrhage | 10072694 |
| Chronic pigmented purpura | 10072726 |
| Iliac artery rupture | 10072789 |
| Chance fracture | 10073162 |
| Brain stem haematoma | 10073230 |
| Penile contusion | 10073352 |
| Post procedural contusion | 10073353 |
| Eye contusion | 10073354 |
| Genital contusion | 10073355 |
| Cardiac contusion | 10073356 |
| Spleen contusion | 10073533 |
| Spinal subdural haemorrhage | 10073563 |
| Spinal subarachnoid haemorrhage | 10073564 |
| Bone marrow haemorrhage | 10073581 |
| Instillation site haematoma | 10073609 |
| Instillation site haemorrhage | 10073610 |





| PT Term | Code |
|---------------------------------------------------------|----------|
| Instillation site bruise | 10073630 |
| Epidural haemorrhage | 10073681 |
| Haemophilic pseudotumour | 10073770 |
| Osteochondral fracture | 10073853 |
| Neonatal gastrointestinal haemorrhage | 10074159 |
| Lymph node haemorrhage | 10074270 |
| Sacroiliac fracture | 10074362 |
| Gastrointestinal polyp haemorrhage | 10074437 |
| Traumatic haemothorax | 10074487 |
| Stoma site haemorrhage | 10074508 |
| Limb fracture | 10074551 |
| Spontaneous haemorrhage | 10074557 |
| Deep dissecting haematoma | 10074718 |
| Hyperfibrinolysis | 10074737 |
| Oral mucosa haematoma | 10074779 |
| Spinal fusion fracture | 10074807 |
| Arterial intramural haematoma | 10074971 |
| Eyelid contusion | 10075018 |
| Nasal septum haematoma | 10075027 |
| Administration site bruise | 10075094 |
| Administration site haematoma | 10075100 |
| Administration site haemorrhage | 10075101 |
| Internal haemorrhage | 10075192 |
| Activated partial thromboplastin time ratio abnormal | 10075284 |
| Activated partial thromboplastin time ratio fluctuation | 10075286 |
| Activated partial thromboplastin time ratio increased | 10075287 |
| Aponeurosis contusion | 10075330 |
| Cerebral aneurysm perforation | 10075394 |
| Grey Turner's sign | 10075426 |
| Medical device site bruise | 10075570 |
| Medical device site haematoma | 10075577 |
| Medical device site haemorrhage | 10075578 |
| Acute haemorrhagic ulcerative colitis | 10075634 |
| Carotid artery perforation | 10075728 |
| Aortic perforation | 10075729 |
| Lower limb artery perforation | 10075730 |
| Iliac artery perforation | 10075731 |
| Arterial perforation | 10075732 |





| PT Term | Code |
|---------------------------------------------|----------|
| Venous perforation | 10075733 |
| Cerebral artery perforation | 10075734 |
| Vertebral artery perforation | 10075735 |
| Basilar artery perforation | 10075736 |
| Renal artery perforation | 10075737 |
| Splenic artery perforation | 10075738 |
| Femoral artery perforation | 10075739 |
| Subclavian artery perforation | 10075740 |
| Superior vena cava perforation | 10075741 |
| Inferior vena cava perforation | 10075742 |
| Subclavian vein perforation | 10075743 |
| Iliac vein perforation | 10075744 |
| Femoral vein perforation | 10075745 |
| Mucocutaneous haemorrhage | 10076048 |
| Spinal cord haematoma | 10076051 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Oral blood blister | 10076590 |
| Chest wall haematoma | 10076597 |
| Subarachnoid haematoma | 10076701 |
| Periventricular haemorrhage neonatal | 10076706 |
| Basal ganglia haematoma | 10077031 |
| Vein rupture | 10077110 |
| Surgical fixation of rib fracture | 10077270 |
| Periosteal haematoma | 10077341 |
| Haemorrhagic breast cyst | 10077443 |
| Oesophageal intramural haematoma | 10077486 |
| Vascular access site haemorrhage | 10077643 |
| Vascular access site haematoma <sup>a</sup> | 10077647 |
| Vascular access site rupture | 10077652 |
| Joint microhaemorrhage | 10077666 |
| Vascular graft haemorrhage | 10077721 |
| Vascular access site bruising | 10077767 |
| Bursal haematoma | 10077818 |
| Intestinal varices haemorrhage | 10078058 |
| Oral contusion | 10078170 |
| Extra-axial haemorrhage | 10078254 |
| Costal cartilage fracture | 10078358 |
| Lisfranc fracture | 10078749 |





| PT Term | Code |
|-----------------------------------------------------|----------|
| Traumatic intracranial haematoma | 10079013 |
| Retinal aneurysm rupture | 10079121 |
| Bronchial varices haemorrhage | 10079163 |
| Fracture blisters | 10079423 |
| Achenbach syndrome | 10079562 |
| Metaphyseal corner fracture | 10079667 |
| Anal fissure haemorrhage | 10079765 |
| Fracture infection | 10079813 |
| Subchondral insufficiency fracture | 10079864 |
| Eye haematoma | 10079891 |
| Haemorrhagic adrenal infarction | 10079902 |
| Peripheral artery aneurysm rupture | 10079908 |
| Paranasal sinus haemorrhage | 10080108 |
| Pseudofracture | 10080404 |
| Osteophyte fracture | 10080550 |
| Gastrointestinal vascular malformation haemorrhagic | 10080561 |
| Subgaleal haemorrhage | 10080900 |
| Maisonneuve fracture | 10081343 |
| Hypophosphataemic osteomalacia | 10081362 |
| Fothergill sign positive | 10081749 |
| Growth disorder | 10081945 |
| Puncture site haematoma | 10081957 |
| Puncture site bruise | 10082035 |
| Cerebral cyst haemorrhage | 10082099 |
| Pulmonary haemorrhage neonatal | 10082194 |
| Blood loss anaemia | 10082297 |
| Pathological fracture prophylaxis | 10082364 |
| Subendocardial haemorrhage | 10082459 |
| Acquired factor IX deficiency | 10082747 |
| Extradural haematoma evacuation | 10082797 |
| Pathological tooth fracture | 10082930 |
| Pharyngeal contusion | 10083176 |
| Anticoagulant-related nephropathy | 10083346 |
| Urinary bladder haematoma | 10083358 |
| Subcapsular hepatic haematoma | 10083383 |
| Subcapsular splenic haematoma | 10083384 |
| Subcapsular renal haematoma | 10083385 |
| Oral purpura | 10083533 |





| PT Term | Code |
|-----------------------------------------------------|----------|
| Orbital haematoma | 10083565 |
| Spinal fracture treatment | 10083586 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Pancreatic pseudocyst haemorrhage | 10083813 |
| Immune thrombocytopenia | 10083842 |
| Haemangioma rupture | 10084040 |
| Vascular anastomotic haemorrhage | 10084092 |
| Intratumoural haematoma | 10084177 |
| Antiplatelet reversal therapy | 10084904 |
| Urinary occult blood | 10084960 |
| Omental haemorrhage | 10085045 |
| Haemorrhagic occlusive retinal vasculitis | 10085070 |
| Haemorrhagic gastroenteritis | 10085136 |
| Scleral haematoma | 10085163 |
| Jugular vein haemorrhage | 10085298 |
| Gastrointestinal anastomotic haemorrhage | 10085369 |
| Heavy menstrual bleeding | 10085423 |
| Abnormal uterine bleeding | 10085424 |
| Gallbladder haematoma | 10085893 |
| Haemorrhagic cerebellar infarction | 10085944 |
| Peripheral exudative haemorrhagic chorioretinopathy | 10086195 |
| Hypergammaglobulinaemic purpura of Waldenstrom | 10086403 |
| Intracranial haemorrhage neonatal | 10086946 |
| Hepatic artery haemorrhage | 10087132 |

<sup>&</sup>lt;sup>a</sup> The list of PTs in Appendix G was created based on MedDRA Version 25.0; as of MedDRA Version 26.0, LLT Peripheral artery haematoma has been changed from PT Peripheral artery haematoma to PT Vascular access site haematoma.